## STATISTICAL ANALYSIS PLAN (SAP)

**Study Title**: A Double-blind, Randomized-withdrawal, Placebo-controlled Study to Evaluate the Efficacy and Safety of Human Plasma-derived C1-esterase Inhibitor as Add-on to Standard of Care for the Treatment of Refractory Antibody Mediated Rejection in Adult Renal Transplant Recipients

Investigational Medicinal Product: C1-INH (C1-esterase Inhibitor, Human)

Protocol Number: CSL842 3001

Version: FINAL 1.0

Version Date: 10-Dec-2020

**Sponsor:** 

CSL Behring LLC 1020 First Avenue King of Prussia, PA 19406 United States

This document includes information and data that contain trade secrets and privileged or confidential information which is the property of CSL Behring LLC and/or its affiliates ("CSL"). This information must not be made public without written permission from CSL. These restrictions on disclosure will apply equally to all future information supplied to you.

Statistical Analysis Plan

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

# Signature Pages

Authors:

| CSL Behring Study<br>Statistician | Name | Signature | Date (dd/mmm/yyyy) |
|---|---|---|---|
| Author: | PPD | | |
| Title: | PPD | | |
| Company: | CSL Behring LLC | | |

| ESP Lead<br>Statistician | Name | Signature | Date (dd/mmm/yyyy) |
|--------------------------|------|-----------|--------------------|
| Author: | PPD | | |
| Title: | PPD | | |
| Company: | PPD | | |

Statistical Analysis Plan

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

### Approvers:

By signing below, I approve of this version of the Statistical Analysis Plan.

| | Name | Signature | Date (dd/mmm/yyyy) |
|--------------|-----------------|-----------|--------------------|
| Approved by: | PPD | | |
| | , PhD | | |
| Title: | PPD | | |
| Company: | CSL Behring LLC | | |

| | Name | Signature | Date (dd/mmm/yyyy) |
|--------------|-----------------|-----------|--------------------|
| Approved by: | PPD , MD | | |
| Title: | 110 | | |
| Company: | CSL Behring LLC | | |

## **Table of Contents**

| Table of Contents | | 4 |
|------------------------------------|-------------|----|
| List of Tables | | 7 |
| List of Figures | | 8 |
| 1 Modification History | | 9 |
| 2 List of Abbreviations | | 10 |
| • | | |
| , , | ıts | |
| | point | |
| | Endpoints | |
| | • | |
| | d Blinding | |
| 4.5 Determination of the Sample S | Size | 22 |
| 4.6 Planned Interim Analyses and | Reviews | 25 |
| 5 Changes in the Conduct of Plann | ed Analyses | 25 |
| 6 Study Analysis Sets | | 26 |
| 6.1 Screened Analysis Set | | 26 |
| 6.2 Enrolled Analysis Set | | 26 |
| 6.3 Intent-to-Treat Analysis Set | | 26 |
| 6.4 Modified Intent-to-Treat Analy | ysis Set | 27 |
| 6.5 Safety Analysis Sets | | 27 |
| 6.6 Pharmacokinetic Analysis Set | | 27 |
| 6.7 CCI | | |
| 7 General Considerations | | 28 |
| 7.1 Multicenter Studies | | 29 |
| 7.2 Treatment Descriptors | | 29 |

| 7.3 | Multiple Comparisons and Multiplicity | . 29 |
|---|---|---|
| 8 D | ata Handling Conventions | . 30 |
| 8.1 | Missing Data | . 30 |
| 8.1.1 | Imputation of Non-Date Missing Data | . 30 |
| 8.1.2 | Imputation of Partial Dates | |
| 8.2 | Derived Variables | . 33 |
| 8.2.1 | Reference Dates | . 33 |
| 8.2.2 | Study Day for Safety Measures | . 34 |
| 8.2.3 | Study Day for Efficacy | . 34 |
| 8.2.4 | Durations | . 34 |
| 8.2.5 | Baseline Definition. | . 34 |
| 8.2.6 | Change From Baseline | . 35 |
| 8.2.7 | Multiple Assessments | . 35 |
| 8.2.8 | Actual Treatment | . 36 |
| 8.2.9 | Derived Variables | |
| 8.3 | Study Periods Relative to Treatment | . 38 |
| 8.3.1 | Time in Relation to Treatment | . 38 |
| 8.3.2 | Study Time Periods for AEs | . 38 |
| 8.3.3 | Study Time Periods for Prior and Concomitant Medications | . 39 |
| 9 S1 | tudy Population | . 39 |
| 9.1 | Disposition of Subjects | . 39 |
| 9.2 | Protocol Deviations | . 40 |
| 9.3 | Demographic and Baseline Characteristics | . 40 |
| 9.3.1 | Demographics | . 41 |
| 9.3.2 | | . 41 |
| 9.4 | Prior and Concomitant Medications | . 42 |
| 9.5 | Medical History | . 43 |
| 10 E | fficacy | . 43 |
| 10.1 | Analysis of Proportion of Subjects With Loss of Response at the End-of-TP2 | . 43 |
| 10.1.1 | | |
| | | . 44 |
| 10.2 | Analysis of key Secondary Endpoint Proportion of Subjects With All-Cause Allograft Failure Through the Responder Follow-up Period (ie, Within 48 Months After Enrollment) | (4m |
| | rature I nrough the Responder Follow-up Period (le, Within 48 Months After Enrollme | |

| 10.3 | Analysis of Time to All-Cause Allograft Failure Through 48 Months After Enrollment | . 45 |
|---|---|---|
| 10.4 | Analysis of the Change in eGFR From Baseline to End-of-TP1 | . 45 |
| 10.5 | Analysis of Responders at the End-of-TP1 | . 45 |
| 10.6 | Analysis of the Change in eGFR From End-of-TP1 to the End-of-TP2 | . 45 |
| 10.7 | Analysis of the Rate of Change of eGFR in Treatment Period 2 | . 45 |
| 10.8 | CCI | |
| 10.9 | CCI | |
| 10.10 | Analysis of C1-INH Functional Activity | . 46 |
| 10.11 | CCI | |
| 10.12 | Analysis of Plasmapheresis Sessions | . 46 |
| 10.13 | CCI | |
| 10.14 | CCI | |
| 10.15 | CCI | L |
| 10.16 | | |
| 10.17 | CCI | |
| 10.17 | | |
| 10.18 | Trough IVIg Concentrations at Designated Time Points. | . 47 |
| 10.19 | CCI | |
| 10.20 | Treatment Compliance | . 48 |
| 11 S | afety Analyses | . 49 |
| 11.1 | Extent of Exposure | . 49 |
| | Adverse Events | |
| 11.3 | Adverse Events of Special Interest (AESI) | . 51 |
| 11.4 | Deaths and Serious Adverse Events | . 51 |
| 11.5 | Adverse Events Leading to Discontinuation of Study Treatment, Withdrawal from the Study, and Other Significant Adverse Events | 52. |
| 11.6 | Pregnancies | |
| 11.7 | | |
| 11.7.1 | | |
| 11.7.2 | | |

| | _ | | |
|---|---|---|---|
| 11.8 | Other Sa | afety Measures | 53 |
| 11.8.1 | Vital | Signs | 53 |
| 12 Pl | harmacol | cinetics | 53 |
| 12.1 | PK Sam | pling Schedule | 54 |
| 12.2 | Plasma 1 | PK Endpoints | 54 |
| 12.3 | Summar | ry of C1-INH Antigen and Functional Activity Plasma Concentrations | 55 |
| 12.4 | Summar | ry of C1-INH PK Parameters | 55 |
| 12.5 | Pharma | cokinetic Analysis Data Flow | 56 |
| 13 | CI | | |
| 14 | CI | | |
| 15 R | eferences | 3 | 56 |
| 16 A | ppendice | s | 58 |
| 16.1 | | dized MedDRA Query for Embolic and Thrombotic Events (Narrow) (SM | |
| 16.2 | Standard | dized MedDRA Query - Anaphylactic Reaction (Broad) (SMQ Code: 200 | 00021)69 |
| | | List of Tables | |
| Table | 1 | Primary Endpoint | 14 |
| Table | 2 | Secondary Endpoints | 15 |
| Table | 3 | CCI | |
| Table | 4 | Summary of dose and dosing regime | 18 |
| Table | 5 | Description of C1-INH | 20 |
| Table | 6 | Description of Placebo | 21 |

# **List of Figures**

| Figure 1 | Study Overview | 12 |
|---|---|---|
| Figure 2 | Individual variations of eGFR in C1-INH patients | 23 |
| Figure 3 | Stratification of Graft Survival After ABMR Therapy Based on Prognostic Scoring | 25 |

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

# 1 Modification History

| Version | Effective<br>Date | Author of<br>Modification | Reason for Change |
|---|---|---|---|
| 0.2 (misleading<br>version<br>numbering, had<br>been version 1.0) | 21/Jun/2018 | PPD | N/A - First Version |
| 1.0 | 13/Dec/2018 | PPD | Implementation of sponsor comments |
| 2.0 | 27Nov2020 | PPD | Updated document following study<br>termination decision by sponsor |
| 3.0 | 08Dec2020 | PPD | Implementation of sponsor review comments |
| Final 1.0 | 10Dec2020 | PPD | NA |

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

### 2 List of Abbreviations

| ABMR Antibody-Mediated Rejection AE Adverse Event AMR Antibody-mediated Rejection ADAM Analysis Data Model CDISC Clinical Data Interchange Standards Consortium C1-INH C1-esterase Inhibitor Cg Chronic Glomerulopathy CP Conditional Power CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin Col Col FK Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine TEE Thromboembolic Events | Abbreviation | Term |
|---|---|---|
| AMR Antibody-mediated Rejection ADaM Analysis Data Model CDISC Clinical Data Interchange Standards Consortium C1-INH C1-esterase Inhibitor Cg Chronic Glomerulopathy CP Conditional Power CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin SGI GGI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>α</sub> Serum Creatinine | ABMR | Antibody-Mediated Rejection |
| ADaM Analysis Data Model CDISC Clinical Data Interchange Standards Consortium C1-INH C1-esterase Inhibitor Cg Chronic Glomerulopathy CP Conditional Power CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin GCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>ττ</sub> Serum Creatinine | AE | Adverse Event |
| CDISC Clinical Data Interchange Standards Consortium C1-INH C1-esterase Inhibitor Cg Chronic Glomerulopathy CP Conditional Power CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI SCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>C</sub> Serum Creatinine | AMR | Antibody-mediated Rejection |
| C1-INH C1-esterase Inhibitor Cg Chronic Glomerulopathy CP Conditional Power CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scα Serum Creatinine | ADaM | Analysis Data Model |
| Cg Chronic Glomerulopathy CP Conditional Power CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin GCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>α</sub> Serum Creatinine | CDISC | Clinical Data Interchange Standards Consortium |
| CP Conditional Power CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin SCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAF Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | C1-INH | C1-esterase Inhibitor |
| CSL CSL Behring LLC DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI CCI CCI CCI SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | Cg | Chronic Glomerulopathy |
| DGF Delayed Graft Function DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI CCI SCI SCI SCI SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | CP | Conditional Power |
| DSA Donor-specific Antibody DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>Cr</sub> Serum Creatinine | CSL | CSL Behring LLC |
| DVT Deep Vein Thrombosis eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | DGF | Delayed Graft Function |
| eCRF Electronic Case Report Form eGFR Estimated Glomerular Filtration Rate GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin GGI GGI GGI FK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | DSA | Donor-specific Antibody |
| eGFR Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin GGI GCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | DVT | Deep Vein Thrombosis |
| GCP Good Clinical Practice GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI CCI RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>cr</sub> Serum Creatinine | eCRF | Electronic Case Report Form |
| GFR Glomerular Filtration Rate HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>CT</sub> Serum Creatinine | eGFR | |
| HR Hazard Ratio ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>CT</sub> Serum Creatinine | GCP | Good Clinical Practice |
| ICH International Conference on Harmonization IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | GFR | Glomerular Filtration Rate |
| IMP Investigational Medicinal Product IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | HR | Hazard Ratio |
| IDMC Independent Data Monitoring Committee IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | ICH | International Conference on Harmonization |
| IRT Interactive Response Technology ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>α</sub> Serum Creatinine | IMP | Investigational Medicinal Product |
| ITT Intent-to-Treat IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | IDMC | Independent Data Monitoring Committee |
| IV Intravenous IVIg Intravenous Immunoglobulin CCI CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>CT</sub> Serum Creatinine | IRT | Interactive Response Technology |
| IVIg Intravenous Immunoglobulin CCI PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>CT</sub> Serum Creatinine | ITT | Intent-to-Treat |
| PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>C</sub> Serum Creatinine | IV | Intravenous |
| PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>C</sub> Serum Creatinine | | Intravenous Immunoglobulin |
| PK Pharmacokinetic RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>α</sub> Serum Creatinine | | |
| RIS Run-in Safety RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | | |
| RWS Randomized Withdrawal Safety SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous S <sub>C</sub> Serum Creatinine | | Pharmacokinetic |
| SAE Serious Adverse Event SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | RIS | Run-in Safety |
| SAP Statistical Analysis Plan SC Subcutaneous Scr Serum Creatinine | RWS | Randomized Withdrawal Safety |
| SC Subcutaneous S <sub>cr</sub> Serum Creatinine | SAE | Serious Adverse Event |
| S <sub>cr</sub> Serum Creatinine | | Statistical Analysis Plan |
| | SC | Subcutaneous |
| TEE Thromboembolic Events | Sα | Serum Creatinine |
| | TEE | Thromboembolic Events |

### 3 Purpose

This is the statistical analysis plan (SAP) for the Clinical Study Report for study CSL842\_3001. This SAP provides details of the planned statistical analyses of the primary and relevant secondary endpoints for which data are available. This study was terminated by the sponsor on September 15, 2020 for administrative reasons. At the time of termination, 13 subjects were randomized and 2 subjects were still in treatment (1 subject in TP2 and another subject in retreatment). The study database will be locked after the completion of the dosing regimens of these 2 subjects. Based n the termination of the study, many analysis discussed in the protocol will not be able to be performed (for example, all 4 year endpoints are unattainable).

This SAP complies with the International Conference on Harmonisation (ICH) Harmonised Tripartite Guideline Topic E9, Statistical Principles for Clinical Trials. It is based upon the Clinical Study Protocol (dated 01-March-2017) and Study Protocol Amendment Version 1.0 (dated 30-August-2017), Study Protocol Amendment Version 2.0 (dated 23-January 2019), and Study Protocol Amendment Version 3.0 (dated 31-January 2020).

### 4 Study Design

# 4.1 Study Design

Study CSL842\_3001 is a randomized withdrawal, double-blind, placebo-controlled, multi-center study. A schematic of the design is shown in Figure 1. Full details may be found in Section 3 of the Clinical Study Protocol.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)



AMR = antibody-mediated rejection; C1-INH = C1-esterase inhibitor; human; IVIg = intravenous immunoglobulin; MFI = mean fluorescence intensity; TP1 = Treatment Period 1; Treatment Period 2

Note: Post-treatment Follow-up Period is for responders.

- <sup>a</sup> Intravenous immunoglobulin (IVIg) will be administered every 4 weeks to all subjects at a dose of 2 grams/kg. The dose must be administered over a minimum period of at least 2 days, and may be administered over a period of up to 5 days. Plasmapheresis may be administered based on local DSA results and Principal Investigator's judgement.
- <sup>b</sup> Intravenous (IV) C1-INH (60 IU/kg) will be administered to each subject over the first 13 days of TP1 for a total of 5 doses. Thereafter, subcutaneous (SC) C1-INH (60 IU/kg twice weekly) will be administered to each subject for the remainder of TP1.
- c If DSA ≥ 2000 MFI in local lab in TP2 or Retreatment Period, IVIg may be administered to subjects at a dose of 2 grams/kg every 4 weeks. The dose must be administered over a minimum period of at least 2 days, and may be administered over a period of up to 5 days. Plasmapheresis may be administered based on local DSA results and Principal Investigator's judgement (Section 5.4.2 of the protocol).
- <sup>d</sup> During the TP2, eligible subjects will be randomized 1:1 to receive treatment with investigational product (C1-INH [60 IU/kg] or placebo) subcutaneously twice weekly.
- <sup>e</sup> Retreatment Period(s) are blinded and subjects will receive the same investigational product treatment assignment as received during Treatment Period 2.
- <sup>f</sup> Response is defined as an End-of-TP1 eGFR (mean of Week 11 and Week 12 eGFR) that is  $\geq$  20 mL/min/1.73 m<sup>2</sup> and  $\geq$  90% of the baseline eGFR (mean of Screening and the Day 1 eGFR)).
- g AMR Recurrence or persistence in Responder Follow-up Period is proven by biopsy, evidenced by infiltrating neutrophils and/or monocytes with or without the presence of C4d (g > 0, v > 0, and/or ptc > 0 (if C4d is negative,  $g + ptc \ge 2$ , (Section 8.1.3.3 of the protocol).

- During open-label TP1, all eligible subjects will receive treatment with C1-INH (60 IU/kg) in combination with standard of care for 13 weeks. At the conclusion of TP1, subjects who demonstrate a treatment response (see Section 8.2.9) will be randomized to continue in the study in TP2. Subjects who are considered non-responders will enter the Non-responder Follow-up Period during which they will be followed for up to 48 months.
- During the blinded TP2, randomized subjects will either continue treatment with C1-INH (60 IU/kg) or begin treatment with placebo (both in combination with IVIg and plasmapheresis) for 25 weeks, according to the randomization schedule.
- At the conclusion of TP2, randomized subjects will enter the Responder Follow-up Period, where they will be observed for approximately 39 months until Study Month 48.

Randomized subjects who experience a biopsy-proven AMR recurrence or who have persistent AMR during the Responder Follow-up will be permitted to undergo blinded retreatment with either C1-INH or placebo (both in combination with standard of care treatment). Subjects who participate in a Retreatment Period will receive blinded investigational product (C1-INH or placebo) according to their TP2 treatment assignment, in combination with standard of care.

## 4.2 Study Objectives and Endpoints

## 4.2.1 Primary Objective and Endpoint

## 4.2.1.1 Primary Objective

The primary objective of the study is to evaluate the efficacy of C1-INH in the treatment of refractory AMR in renal allograft recipients.

Protocol Number: CSL842\_3001 Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

# 4.2.1.2 Primary Endpoint

Table 1 Primary Endpoint

| Endpoint | Summary Measure |
|---|---|
| Loss-of-response | Proportion of subjects with loss-of-response at the End-of-TP2. |
| during TP2. | Loss-of-response at the End-of-TP2 is defined as any 1 of the following 3 conditions: |
| | • End-of-TP2 eGFR (mean of Week 36 and Week 38 eGFR) that is not stable, defined as: |
| | <ul> <li>End-of-TP2 eGFR that is &lt; 90% of the End-of-TP1<br/>eGFR for subjects whose End-of-TP1 eGFR (mean of<br/>Week 11 and Week 12 eGFR) is ≥ 100% of baseline,</li> </ul> |
| | <ul> <li>End-of-TP2 eGFR that is &lt; 90% of baseline for subjects<br/>whose end-of- TP1 eGFR is ≥ 90% of baseline and<br/>&lt;100% of baseline,</li> </ul> |
| | Allograft failure (defined by allograft nephrectomy, or institution of permanent dialysis, or return to the transplant waitlist for renal transplant, whichever occurs first), |
| | Subject death by any cause. |

eGFR = estimated glomerular filtration rate; TP1= Treatment Period 1; TP2 = Treatment Period 2

# **4.2.1.3** Intended Primary Study Hypothesis

Corresponding to the primary objective, the superiority of C1-INH relative to placebo are measured by the primary endpoint, proportion of subjects with loss of response at the End-of-TP2, based on the Modified Intent-to-Treat analysis. The null hypothesis was to be tested using the Wald statistic derived from maximum likelihood estimation of the logistic model with a Type I error rate of 0.05 (two-sided test). Symbolically, the null and alternative hypotheses are expressed as follows:

 $H_0: \beta_T = 0 \text{ vs } H_1: \beta_T \neq 0$ 

where  $\beta_T$  is the coefficient of treatment in the logistic regression model.

Since the study terminated early, there will be no formal hypothesis testing for any endpoints.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

# 4.2.2 Secondary Objectives and Endpoints

## 4.2.2.1 Secondary Objectives

The secondary objectives of the study are:

- 1. To further evaluate the efficacy of C1-INH in the treatment of refractory AMR in renal allograft recipients.
- 2. To evaluate the safety of C1-INH in the treatment of refractory AMR in renal allograft recipients.
- 3. To evaluate the pharmacokinetics (PK) of C1-INH during the treatment of refractory AMR in renal allograft recipients.

## 4.2.2.2 Secondary Endpoints

**Table 2** Secondary Endpoints

| Secondary<br>Objective | Endpoints | Summary Measure |
|---|---|---|
| 1 All-cause allograft failur through the Responder | allograft failure<br>through the | Proportion of subjects with all-cause allograft failure through the Responder Follow-up Period (ie, within 48 months after enrollment). Allograft failure is defined as 1 of the following: |
| | Follow-up Period | • Allograft nephrectomy, institution of permanent dialysis, or return to the transplant waitlist for renal transplant, whichever occurs first, OR |
| | | • Subject death by any cause. |
| 1 | Change in eGFR from baseline to TP1 | The difference between the End-of-TP1 eGFR and baseline eGFR. |
| 1 | Change in eGFR from TP1 to the End-of -TP2. | The difference between the End-of-TP2 eGFR and the End-of-TP1 eGFR. |
| 1 | The rate of change of eGFR. | The rate of change of eGFR during TP2 as defined by the slope of the mean regression of eGFR over time in TP2. |
| 1 | Time (weeks) to<br>all-cause allograft<br>failure through the<br>Responder<br>Follow-up Period | Time (weeks) to all-cause allograft failure through the Responder Follow-up Period (ie, within 48 months after enrollment). |

| Secondary<br>Objective | Endpoints | Summary Measure |
|---|---|---|
| 1 | Responder status at the End-of-TP1. | Proportion of responders at the End-of-TP1. Response is defined as End-of-TP1 eGFR that is $\geq 20$ mL/min/1.73 m <sup>2</sup> and $\geq 90\%$ of the baseline eGFR. |
| 1 | Subject death through the Responder Follow-up Period. | Proportion of subjects surviving through the Responder Follow-up Period. |
| 2 | Any AE assessed as related to investigational product during TP1 and during TP2. | Proportion of subjects with any AE assessed as related to investigational product. |
| 3 | Pre-dose C1-<br>esterase inhibitor<br>functional activity<br>at Day 1, Week<br>12, and Week 38. | Mean pre-dose C1-esterase inhibitor functional activity at Day 1, Week 12, and Week 38. |
| 3 | For the subset of subjects with sequential PK sampling, C1-esterase inhibitor functional activity C <sub>max</sub> , and AUC <sub>0-t</sub> after IV and/or SC administration of C1-INH. | C1-esterase inhibitor functional activity $C_{max}$ and $AUC_{0-t}$ for IV and SC administration. |

AE = adverse event; AUC<sub>0-t</sub> = area under the plasma-concentration time curve 0 to a definite time; C<sub>max</sub> = maximum concentration; eGFR = estimated glomerular filtration rate; IV = intravenous; PK = pharmacokinetic; SC = subcutaneous; TP1 = Treatment Period 1; TP2 = Treatment Period 2

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

4.2.2.3 <sup>CCI</sup>



4.2.2.4 CCI





### 4.3 Study Treatments

#### Dose and Dosing Regimen

A summary of dose and dosing regimen is shown in Table 4.

Table 4 Summary of dose and dosing regime

| Timeframe | Intravenous<br>Administration | Subcutaneous<br>Administration |
|---|---|---|
| Treatment Period 1: The Day 1 Visit to the Day 13 Visit <sup>a</sup> | 60 IU/kg C1-INH | Not applicable |
| Treatment Period 1: The Day 14 Visit to the Week 12 2nd Visita | Not Applicable | 60 IU/kg C1-INH |
| Treatment Period 2: Week 13 to the Week 38 Visit <sup>b</sup> | Not Applicable | 60 IU/kg C1-INH<br>OR<br>0.12 mL/kg Placebo |
| Re-treatment Period: The Retreatment Day 1 Visit to<br>the Retreatment Week 26 Visit.c | Not Applicable | 60 IU/kg C1-INH<br>OR<br>0.12 mL/kg Placebo |

IV = intravenous; SC = subcutaneous

Note: Week 13 is the final visit of Treatment Period 1 for non-responders and the first visit of Treatment Period 2 for responders.

Treatment Period 1 is open-label and each subject will receive C1-INH. C1-INH (60 IU/kg) will be administered IV to each subject over the first 13 days of Treatment Period 1 for a total of 5 doses. Thereafter, C1-INH (60 IU/kg twice weekly) will be administered SC to each subjects for the remainder of Treatment Period 1. The first dose of randomized investigational product will be administered to responders at the Week 13 Visit.

b Treatment Period 2 is blinded and subjects will be randomized 1:1 to treatment with investigational product (C1-INH [60 IU/kg] or placebo) subcutaneously twice weekly.

<sup>&</sup>lt;sup>c</sup> Retreatment Period(s) are blinded and subjects will receive the same investigational product treatment assignment as received during Treatment Period 2.

### **Treatment Period 1**

C1-INH will be administered to all subjects during Treatment Period 1 in an open-label manner. Five doses of C1-INH will be administered intravenously to subjects at the Day 1, 4, 7, 10, and 13 Visits. Intravenous C1-INH will be administered at the study site during site visits. Subcutaneous C1-INH will be administered every 3 to 4 days (ie, twice weekly) beginning at the Day 14 Visit and for the remainder of Treatment Period 1. Subcutaneous C1-INH is required to be administered at the study site during site visits, but at other times may instead be administered at home by a medical professional ((eg, a home visit nurse) or by the subject under the supervision of a medical professional.

#### **Treatment Period 2**

Investigational product (ie, C1-INH or placebo) will be administered to all subjects during Treatment Period 2 in a double-blind manner. Subcutaneous investigational product will be administered every 3 to 4 days (ie, twice weekly) during Treatment Period 2. Subcutaneous C1-INH is required to be administered at the study site during site visits, but at other times may instead be administered at home by a medical professional (eg, a home visit nurse) or by the subject under the supervision of a medical professional.

#### Retreatment Period

Subjects may undergo retreatment during the Responder Follow-up Period with the blinded investigational product to which they were randomized in TP2. Retreatment may occur following a diagnosis of recurrent or persistent AMR by biopsy, evidenced by infiltrating neutrophils and/or monocytes with or without the presence of C4d (glomerulitis [g] > 0, intimal arteritis [v] > 0, and/or peritubular capillaritis [ptc] > 0; if C4d is negative,  $g+ptc \ge 2$ ). Retreatment may start at any time during the Responder Follow-up Period, and will last for 26 weeks or until the Month 48 Visit, whichever occurs first. The Retreatment Period may also be shorter than 26 weeks at the investigator's discretion.

During the Retreatment Period, SC investigational product will be administered twice weekly (approximately every 3 to 4 days). During the Retreatment Period (if needed), SC C1-INH will be administered either at the site or may be dispensed to the subject and administered SC at home either by a medical professional or by the subject under the supervision of a medical professional.

### Subcutaneous Administration of the Investigational Product

Subcutaneous administration of the investigational product should be via a single SC injection in the abdomen, thigh, upper arm, or other appropriate location. The twice weekly administration of investigational product beginning at the Day 14 Visit and during any Retreatment Period (if applicable). The suggested interval between each administration of investigational product is 3 or 4 days (ie, twice weekly). In addition, the investigational product should ideally be administered at approximately the same time on each day. A missed injection should be administered as soon as possible, unless within 24 hours of the next scheduled injection; in this situation, the missed injection should be omitted, and the administration of investigational product should occur at the next scheduled day and time. The volume of investigational product to be administered will be based on each subject's body weight (from the Screening physical examination) and will not be adjusted during the study.

#### **Description of Investigational Products**

The investigational products for this study are C1-INH and placebo. A description of C1-INH and Placebo and given in Table 5 and Table 6 respectively.

Table 5 Description of C1-INH

| Substance name | C1-esterase Inhibitor, Human (500 IU/mL) |
|---|---|
| Active substance | C1-esterase inhibitor (human) |
| Trade name | Not applicable |
| Dosage form | Lyophilized powder for reconstitution; 1500 IU C1-INH per single-use vial. |
| Dose | 60 IU/kg |
| Mode of administration | Intravenous / subcutaneous injection |

Before use, each vial of C1-INH is reconstituted with 3 mL water for injection. 60 IU/kg C1-INH is equivalent to a volume of 0.12 mL/kg.

Statistical Analysis Plan

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

Table 6Description of Placebo

| Substance number | Not applicable |
|---|---|
| Substance | Excipients of C1-INH plus albumin |
| Trade name Not applicable | |
| Dosage form Lyophilized powder for reconstitution | |
| Dose | 0.12 mL/kg |
| Mode of administration | Subcutaneous injection |

Before use, each vial of placebo is reconstituted with 3 mL water for injection.

The volume of placebo will be based on the body weight obtained with vital signs assessment at the Screening Visit, and will not be changed through the study. The actual dose of placebo will be rounded to the lowest 1 mL as if the subject receiving C1-INH.

### 4.4 Randomization Procedures and Blinding

#### **Randomization Procedures**

All subjects will receive open-label C1-INH during Treatment Period 1. Subjects who are eligible for Treatment Period 2 will be assigned to either continued C1-INH or matched placebo in accordance with a computer-generated randomization list. Investigational product assigned in Treatment Period 2 will be allocated on a 1:1 ratio. The randomization will be stratified on the following 2 factors:

- Donor Specific Antibodies (DSA): sensitized prior to transplantation versus de novo. De novo is defined as the development of DSA after transplantation. In the case of both sensitized and de novo, the subject will be considered sensitized for stratification purposes.
- AMR severity: severe versus non-severe (ie all other severities). Severe AMR is defined as new onset oliguria (< 400 cc / 24 hours) or anuria with the current episode of AMR.

Therefore, there will be a total of 4 strata (2 factors, 2 levels per factor). The randomization will be permuted block within each stratum. Treatment assignment will be determined centrally. The randomization list will be generated and managed by the study's interactive response technology (IRT) external service provider.

The study database will be locked once all the randomized subjects currently in the study complete week 38 visit and re-treatment period as described in Section 3. The study will be unblinded for final analysis of the primary efficacy endpoint.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

### **Maintaining the Blind**

Treatment Period 1 is open-label. Treatment Period 2 is double-blind. During Treatment Period 2, the blind will be maintained for investigational site staff, including investigators, subjects, and CSL.

### **Emergency Unblinding**

In emergency situations involving the safety of the subject, the investigator may break the blind using the IRT system. The reason for unblinding the randomization code must be fully documented. Emergency unblinding will be performed using the IRT. Steps for navigating the IRT for emergency unblinding are defined in the IRT manual.

## 4.5 Determination of the Sample Size

#### Sample Size Based on the Primary Efficacy Endpoint

The sample size is based on the primary efficacy endpoint of loss-of-response status (binary endpoint of loss-of-response or not), at the End-of-TP2 (ie, within 25 weeks after randomization). The null hypothesis is that there is no difference between C1-INH and placebo with respect to the proportion of subjects with loss-of-response at the End-of-TP2. Let  $p_0$  and  $p_1$  be the expected proportion of subjects with loss-of-response in TP2 in the placebo and C1-INH treatment groups, respectively. The alternative is that there is a difference between the treatment groups. That is,  $H_0$ :  $p_0 = p_1$  versus  $H_1$ :  $p_0 \neq p_1$ .

The power procedure in SAS STAT software (Cary, NC SAS Institute Inc.) was used to estimate the sample size, based on the likelihood ratio chi-square test. Determination of the sample size was based on the following assumptions:

- The proportions of subjects experiencing loss-of-response at the End-of-TP2 will be 0.75 with placebo and 0.30 with C1-INH.
- There will be at least 90% power to detect a statistically significant effect with two-sided test with alpha = 0.05.
- Logistic regression model with treatment effect will be used for the primary efficacy analysis. Wald test statistic for treatment effect from Logistic regression has approximately same distribution as chi-square [Fleiss et al, 2003]. Therefore, the sample size calculation based on chi-square test is used to ensure similar power for hypothesis testing.
- Treatment allocation will be 1:1.

• The planned interim analysis for futility will not impact the type 1 error for the final analysis. Under these assumptions, a total of 60 subjects (30 randomized to C1-INH and 30 randomized to placebo) will provide approximately 95% power. The study was planned to enroll a sufficient number of subjects (up to 175) to ensure that 60 subjects are randomized.

The assumptions above are based on a prospective single-arm pilot study to investigate the C1- INH added to high-dose IVIG for the treatment of acute AMR non-responsive to conventional therapy [Viglietti et al, 2016a]. A total of 6 subjects received C1-INH and IVIg for 6 months. The primary endpoint was change in eGFR. These were compared to a historical control of 21 subjects who received IVIg. In the prospectively treated C1-INH group, 0/6 subjects experienced decline in eGFR at 6 months (0; 95% confidence interval [CI], 0 to 46%); and 4/6 subjects had a greater than 20% increase in eGFR (67%; 95% CI, 22% to 96%). In the historical control group, 15/21 subjects (71%; 95% CI, 48% to 89%) experienced decline in eGFR during a comparable 6-month period. The results are presented in Figure 2.

Figure 2 Individual variations of eGFR in C1-INH patients



Left: Distributions of eGFR at time of initial diagnosis (M-3), at the end of first line treatment (SOC; M0) and at the end of C1-INH treatment (M+6) in 6 patients. Right: Individual variations in eGFR between M0 and M+6 in C1-INH patients (green) and historical controls (red). From Viglietti et al. (Viglietti et al., 2016b)

### Power for the analysis of all-cause allograft failure

Allograft survival status (or all-cause allograft failure) at the end of 48 months after enrollment represents clinical confirmation of the effect on the allograft of improving eGFR.

The primary comparison of the proportion of subjects with allograft survival will be between the subjects randomized to placebo or C1-INH. It is anticipated that very few subjects will be lost to follow-up as standard of care mandates close follow up by the transplanting center. This endpoint will be analyzed after all subjects have been followed for 4 years after enrollment.

The power for hypothesis testing of this endpoint was estimated using the power procedure in SAS STAT under the following assumptions:

- The proportions of subjects with allografts surviving at 4 years after enrollment will be 0.25 with the placebo cohort and 0.75 in the C1-INH cohort.
- Alpha = 0.05 (two-sided test).
- Logistic regression model with treatment effect will be used for the primary efficacy analysis. Wald test statistic for treatment effect from Logistic regression has approximately same distribution as chi-square [Fleiss et al, 2003]. Therefore, the sample size calculation based on chi-square test is used to ensure similar power for hypothesis testing.
- Approximately 30 subjects in each randomized treatment groups.

There is greater than 90% power to detect the specified target difference between C1-INH and placebo groups based on sample size of 60 (approximately 30 in the C1-INH cohort and approximately 30 in the placebo cohort).

The 4-year graft survival for placebo of 25% is based on data presented at the American Transplant Congress in Boston [Viglietti et al, 2016b], as shown in Figure 3. This study involved follow-up of kidney transplant recipients with biopsy-proven active AMR diagnosed between 2007 and 2013. Among the subjects who have not responded to standard of care, the 4-year graft survival ranged from approximately 10% to 40% for subjects with high and intermediate risk scores, respectively. The 4-year graft survival for C1-INH of 75% represents what would be expected for subjects who are successfully treated.

Protocol Number: CSL842\_3001 Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

Figure 3 Stratification of Graft Survival After ABMR Therapy Based on Prognostic Scoring





Source: Viglietti et al, 2016b American Transplant Congress Abstract #198

## 4.6 Planned Interim Analyses and Reviews

The study will be monitored by an Independent Data Monitoring Committee (IDMC). The meeting frequency, specific responsibilities, and composition of the IDMC will be outlined in a separate document, the IDMC charter.

The study was terminated by the sponsor on 15 September 2020, therefore, no interim analysis will be conducted.

# 5 Changes in the Conduct of Planned Analyses

There are changes in the planned analyses (from those specified in the protocol) following the sponsor's decision to terminate the study. There will be no analysis of the endpoints below Data from these endpoints will be presented only in subject listings.:

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

- Secondary endpoint of proportion of subjects with all-cause allograft failure through the Responder Follow-up Period,
- Time to all-cause allograft failure through 48 months after enrollment,
- Change in eGFR from End-of-TP1 to the End-of-TP2,
- Rate of change of eGFR in Treatment Period 2,
- CCI
- Plasmapheresis sessions,
- CCI ,
- ,
- Trough IVIg concentrations at designated time points,
- CCI

For other endpoints the statistical analysis was reduced as described in the sections of this SAP.

### 6 Study Analysis Sets

### 6.1 Screened Analysis Set

The Screened analysis will comprise all subjects who provided written informed consent and who underwent study screening procedures.

### 6.2 Enrolled Analysis Set

The Enrolled Analysis Set will comprise all subjects in the Screened Analysis Set who did not fail screening.

#### 6.3 Intent-to-Treat Analysis Set

The Intent-to-Treat (ITT) analysis will comprise all subjects who were randomized. Subjects will be classified according to the investigational product to which they were assigned (ie, continued C1-INH or placebo) regardless of what was actually received. This will be the primary analysis

Protocol Number: CSL842\_3001 Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

set for the analysis of efficacy data. Any subject who received a randomization identification number will be considered to have been randomized.

### 6.4 Modified Intent-to-Treat Analysis Set

All subjects randomized under the original protocol and under all protocol amendments will be included in the Modified ITT (mITT) population except the subjects randomized prior to Amendment 3 who did not satisfy the eligibility criteria updated in Amendment 3. The mITT Analysis Set will be the primary analysis set for the analysis of efficacy data.

## 6.5 Safety Analysis Sets

#### Run-in Safety Analysis Set

The Run-in Safety (RiS) Analysis Set will comprise all subjects who received at least one dose of C1-INH during Treatment Period 1.

#### Randomized Withdrawal Safety Analysis Set

The Randomized Withdrawal Safety (RWS) Analysis Set will include all subjects in the ITT Analysis Set who received at least one dose of the investigational product after randomization during Treatment Period 2. The RWS Analysis Set will be based on the investigational product actually received (ie, continued C1-INH or placebo) during Treatment Period 2. If a C1-INH treatment subject receives one or two doses of placebo and then this is corrected for all subsequent doses they will be classified in the C1-INH treatment group.

## 6.6 Pharmacokinetic Analysis Set

The Pharmacokinetic (PK) Analysis Set will comprise all subjects who received  $\geq 1$  dose of C1-INH and who have  $\geq 1$  measurable level of C1-INH functional activity or C1-INH antigen concentration.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)



#### 7 General Considerations

Analysis datasets will be created according to CDISC standards, and data will be displayed according to reporting standards in this SAP and tables, figures and listings (TFL) formats.

SAS version 9.3 or higher will be used to perform all data analyses and to generate TFLs.

All ICH required data in the database will be presented in data listings.

Continuous variables will be summarized in terms of the number of observations, mean, standard deviation, median, Q1, Q3, minimum and maximum. Other descriptive statistics (eg, quartiles, coefficient of variation) may be reported when appropriate. Categorical variables will be summarized using frequency counts and percentages. Analyses that use other descriptive statistics will have the specific descriptive statistics required identified with the analysis in the applicable SAP section.

All listings will include subject number, treatment group. The laboratory normal reference ranges will be provided and clinical laboratory test results outside the normal reference range will be flagged in the laboratory data listings.

Summary statistics of central tendency will be reported to one more decimal place than the collected data. Summary statistics of variability will be reported to one more decimal place than the commensurate measure of central tendency. For example, the mean and median for age will be reported to one decimal place because it is collected in full years. The standard deviation of age will then be reported to 2 decimal places.

Formatting for dates and times will be: descriptive percentages and proportions will be displayed to one decimal place. Percentages and proportions to be tested will be calculated to 4 decimal places. Durations for events will be display to 1 decimal place.

- Dates only ddmmmyyyy
- Times only hh:mm or hh:mm.ss
- Dates and times ddmmmyyyy hh:mm or ddmmmyyyy hh:mm:ss

In general, only scheduled visits will be included in by-visit summaries. However, worst-case or best-case values (as appropriate) will be derived using both scheduled and unscheduled visits. In general, assessment windows will not be defined for the purpose of classifying measurements obtained outside scheduled assessment times, other than those indicated in the Schedule of Assessments. However, exceptions may apply for creatinine / eGFR.

Actual rather than planned sampling times will be used in the derivation of PK parameters and in the individual concentration-time plots and listing of PK concentration data. Planned times will be used in the descriptive summaries and in mean and median plots. Concentration-time data will be listed according to actual sampling times relative to dosing time.

Deviations from the analyses in this SAP will be identified in the CSR.

#### 7.1 Multicenter Studies

Data from all participating sites will be pooled prior to analysis.

### 7.2 Treatment Descriptors

The following treatment group descriptor will be used on all applicable displays:

| Treatment Group | | Order of Treatment<br>Groups |
|-----------------|-------------|------------------------------|
| Code | Description | |
| A | Placebo | 1 |
| В | C1-INH | 2 |

## 7.3 Multiple Comparisons and Multiplicity

No formal hypothesis testing is planned due to small number of subjects randomized in this study when the study was terminated by the sponsor. Hence multiplicity is not applicable.

## 8 Data Handling Conventions

### 8.1 Missing Data

Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument. These data will be indicated by the use of a "blank" in subject listing displays. Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such provided in the collection instrument.

### 8.1.1 Imputation of Non-Date Missing Data

#### **Non-date Clinical Data**

All available data will be analyzed using suitable statistical methods. For analysis of percent responders, all subjects in the appropriate analysis set (ITT Analysis Set or mITT Analysis Set) will be included in the denominator when calculating the percentages; any subject who drops out of the study at any time after randomization will be defined for the purpose of analysis as a non-responder.

Subjects with the designation of treatment relationship for adverse events (AEs) and serious adverse events (SAEs) missing will have the worst case assumed to impute the relationship: if relationship to study treatment is missing it will be assumed to be "Yes".

In summaries of absolute values and change from baseline, subjects with missing baseline values will not be included in baseline rows or in the change from baseline summary statistics.

# 8.1.2 Imputation of Partial Dates

Imputed dates will not be used to derive study day, duration (eg, duration of adverse events), or elapsed time variables. In addition, imputed dates are not used for deriving the last contact date for overall survival. Imputed dates will be displayed in listings and identified as imputed.

Partial date imputation will follow Analysis Data Model (ADaM) conventions. The ADaM approach is to populate the numeric date variables with the imputed date and add a flag variable to the dataset that indicates the level of imputation.

The flag variable can contain the values: blank, 'D', 'M', 'Y'.

blank: indicates that no imputation was done

D = 'Day': indicates that the day portion of the date is imputed

M = 'Month': indicates that the month and day portions of the date are imputed

Y = 'Year': indicates that the entire date (year, month, and day) is imputed

Algorithms for imputing partial dates for AE and concomitant medications are below.

Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings. They will not be used to calculate duration of AEs. If an AE start or end date is missing, then the duration of the AE will be set to missing.

#### **Adverse Events**

Impute start and end dates for use to derive the reference variables for adverse event start relative to treatment; include any imputed dates in analysis datasets with an identifier as imputed. The reference variables will be used to differentiate as Before-therapy, On-Therapy and Follow-up for AEs (see Section 8.3.2).

| Date | Missing Element | Rule |
|---|---|---|
| Start Date | day, month, and year | Do not impute completely missing AE start dates, AE will be assumed as treatment emergent |
| | day and month | <ul> <li>If the onset year is after the year of the first dose of study drug, then the AE is treatment-emergent.</li> <li>If the onset year is the same as the year of the first dose of study drug and the end date is not before the first dose of study drug, then the AE is treatment-emergent.</li> <li>If the onset year is the same as the year of the first dose of study drug and the end date is before the first dose of study drug, then the AE is not treatment-emergent.</li> <li>If the onset year is before the year of the first dose of study drug, then the AE is not treatment-emergent.</li> </ul> |

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

| Date | Missing Element | Rule |
|---|---|---|
| | day only | <ul> <li>If the start yyyy-mm is after the yyyy-mm of first dose of study drug, then the AE is treatment-emergent.</li> <li>If the start yyyy-mm is the same as the yyyy-mm of the first dose of study drug and the end date is not before the first dose of study drug, then the AE is treatment-emergent.</li> <li>If the start yyyy-mm is the same as the yyyy-mm of the first dose of study drug and the end date is before the first dose of study drug, then the AE is not treatment-emergent.</li> <li>If the onset yyyy-mm is before the yyyy-mm of the first dose of study drug, then the AE is not treatment-emergent.</li> </ul> |
| End Date | any date element | No imputation for completely or partially missing AE end dates; as applicable, report the AE as ongoing and the AE duration as missing. |

### **Concomitant Medication**

Impute start and end dates for use to derive the reference variables for concomitant medication start and end relative to treatment; include any imputed dates in analysis datasets with an identifier as imputed. The reference variables will be used to differentiate before, during and after treatment for the concomitant medication.

| Date | Missing Element | Rule |
|---|---|---|
| Start Date | day, month, and year | Do not impute completely missing concomitant medication start dates. |
| | day and month | <ul> <li>If the onset year is after the year of the first dose of study drug, then the CM is concomitant.</li> <li>If the onset year is the same as the year of the first dose of study drug and the end date is not before the first dose of study drug, then the CM is concomitant.</li> <li>If the onset year is the same as the year of the first dose of study drug and the end date is before the first dose of study drug, then the CM is prior.</li> <li>If the onset year is before the year of the first dose of study drug, then the CM is prior.</li> </ul> |

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

| Date | Missing Element | Rule |
|---|---|---|
| | day only | If the start yyyy-mm is after the yyyy-mm of first dose of study drug, then the CM is concomitant. |
| | | • If the start yyyy-mm is the same as the yyyy-mm of the first dose of study drug and the end date is not before the first dose of study drug, then the CM is concomitant. |
| | | • If the start yyyy-mm is the same as the yyyy-mm of the first dose of study drug and the end date is before the first dose of study drug, then the CM is prior. |
| | | • If the onset yyyy-mm is before the yyyy-mm of the first dose of study drug, then the CM is prior. |

#### **Date of Birth**

Imputation for birth date is only needed if age is missing on eCRF and needs to be recalculated. An incomplete birth date will be imputed as follows:

If only the day is missing – the missing day will be imputed as 15th of the month.

If day and month is missing – missing day and month will be imputed by 1st of July.

A completely missing birth date will not be imputed.

#### 8.2 Derived Variables

The following sections provide a general description of the derived variables for data analyses.

### **8.2.1** Reference Dates

Reference dates are used to assign study periods relative to treatment.

There are three reference dates:

- Because age is an eligibility requirement, the reference date for age is the date of screening.
- The safety reference date is the date of first C1-INH dosing in Treatment Period 1 and will be used to calculate study day for safety measures.
- The reference date for efficacy endpoints is the date of first intake of randomized study treatment in Treatment Period 2 and will be used to calculate study day for efficacy measures.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

## 8.2.2 Study Day for Safety Measures

If the date of interest occurs on or after the safety reference date, then the safety study day will be calculated as (date of interest - safety reference date) + 1. If the date of interest occurs before the safety reference date, then the safety study day will be calculated as (date of interest – safety reference date). There is no safety study day 0.

### 8.2.3 Study Day for Efficacy

The study day for efficacy will be calculated in the same manner as the study day for safety measures but will consider the reference date for efficacy. There is no efficacy Study Day 0.

### **Timings for safety events and interventions**

Safety events and interventions will be classified as follows:

**Before-treatment:** Date is strictly prior to the first administration of open-label C1-INH.

**Treatment-emergent or On-Treatment:** Date is between the first administration of open-label C1-INH and 30 days after the investigational product stop date.

**Post-treatment**: Date is strictly more than 30 days after the investigational product stop date.

#### 8.2.4 Durations

Durations (eg, the duration of an adverse event) and elapsed time will be calculated in days using the SAS DATDIF function.

When reporting durations which are calculated in months, divide the number of days by 30.4375; to report in weeks divide the number of days by 7; to report in years divide the number of days by 365.25. These algorithms for time to event return decimal numbers, and ignore the actual numbers of days in the months or years between start date and stop date. The "year" used in these algorithms is 365.25 days long, and the "month" is one twelfth of that year.

#### **8.2.5** Baseline Definition

Baseline for non-laboratory and laboratory data (except creatinine for eGFR) is defined as the most recent, non-missing value prior to or on the first study treatment dose date/time in Treatment Period 1 (for non-laboratory it is referred to eCRF data and for laboratory data it is referred to local laboratory data).

For subjects who did not receive study treatment during the study, a baseline value will not be calculated. The most recent, non-missing value prior to or on the study treatment dose date / time is based on scheduled assessments only.

Baseline eGFR has been defined as follows in original protocol and amendments:

- For subjects randomized prior to Protocol Amendment 1, dated November 28, 2017, the nadir (minimum) of the eGFR values from screening and Day 1 will be used as the baseline.
- For subjects randomized after Protocol Amendment 1 the mean of the screening and Day 1 values will be used as the baseline.

For the purpose of analysis, baseline eGFR is defined as the mean of the screening and Day 1 values.

Note that a set of vital signs or laboratory values may have different dates for baseline values.

### 8.2.6 Change From Baseline

Change from baseline will only be calculated for measures that have post-baseline records. Change from baseline will be calculated as:

• visit value – baseline value.

Percentage change from baseline will be calculated as:

• (change from baseline / baseline value) \* 100

## **8.2.7** Multiple Assessments

All data will be reported according to the nominal visit date/time for which it was assessed (that is, no visit windows will be applied during dataset creation).

If multiple assessments for the same visit occur, it will be distinguished why this is the case. If a laboratory sample was repeated due to technical problems the results from the valid sample(s) for this visit – the non-missing results – will be used in the analysis. If a laboratory sample was repeated as safety follow-up to monitor abnormal values of the initial sample, the initial sample (revealing the abnormal values) of this visit will be used in the analysis.

Data from all assessments (scheduled and unscheduled), including multiple assessments, will be included in listings.

### 8.2.8 Actual Treatment

The subjects' actual treatment will be derived from exposure data. If a subject's actual treatment is the same as the assigned treatment, then actual treatment is the assigned treatment. If a subject receives a study treatment that is different from the assigned treatment for the entire time of treatment, then actual treatment is the different treatment (the treatment actually received).

#### 8.2.9 Derived Variables

#### **Start and End of Retreatment Periods**

Neither the start and end date of optional Retreatment Period(s) nor the number of individual Retreatment Period(s) will be explicitly recorded in the eCRF. So, the start date of a Retreatment Period will be derived by using the visit date associated with the label of first visit in a Retreatment Period, ie using a visit label of "RT – Day 1 (x)", x – counter of individual Retreatment Period. The end date of a Retreatment Period will be derived in the same way by using the last available date in a chronological order of visit labels in a Retreatment Period, ie using a visit label of "RT – Day 182 (x)", x – counter of individual Retreatment Period. The individual number of Retreatment Period will be derived from the counter (in brackets) given in the visit label of Retreatment Periods.

For analysis purpose, a Retreatment Period will start with the first documented study drug intake on or after first retreatment visit which was identified via the visit label. The end of the Retreatment Period will be identified in a similar way. It will be the last intake of study drug before or on the last retreatment visit which was identified via the visit label.

#### **Demographics**

#### Years of Age

Years of age will be derived as the number of complete years between a subject's birth date and the date of informed consent.

#### **Body mass index**

Body mass index (BMI) will be derived using the following formula:

BMI 
$$(kg/m^2)$$
 = Weight  $(kg) / [Height (m)]^2$
The height at Screening and the dry weight obtained from the medical history will be used. If the dry weight is missing, the weight at Screening will be used. If the weight at Screening is missing, the Day 1 weight will be used.

#### **Efficacy**

#### **Estimated glomerular filtration rate (eGFR)**

eGFR will be derived using the following MDRD formula [Levey et al, 2008]:

eGFR (mL/min/1.73m<sup>2</sup>) = [(175) x (standardized 
$$S_{cr}^{-1.154}$$
) x (age<sup>-0.203</sup>) x (1.212, if black) x (0.742, if female)]

The serum creatinine  $(S_{cr})$  is expressed as mg/dL. The years of age will be derived based on the subject birth date and the date that the  $S_{cr}$  sample was taken.

#### eGFR at the End of Treatment Period 1 (End-of-TP1)

The mean of Week 11 and Week 12 eGFR measurements. If one of the measurements is missing it is then the non-missing value.

#### eGFR at the End of Treatment Period 2 (End-of-TP2)

The mean of Week 36 and Week 38 eGFR measurements. If one of the measurements is missing it is then the non-missing value.

#### Response to Open-Label C1-INH at End of Treatment Period 1 (End-of-TP1)

Responders are defined as subjects whose End-of-TP1 (the mean of Week 11 and Week 12) eGFR  $\geq$  90% of baseline and  $\geq$  20 mL/min/1.73 m<sup>2</sup>. The baseline eGFR is defined as the mean of the screening and Day 1 values in Section 8.2.5.

#### **Loss of Response During Treatment Period 2**

Loss-of-response at the End-of-TP2 is defined as any 1 of the following 3 conditions:

- End-of-TP2 eGFR (mean of Week 36 and Week 38 eGFR) that is not stable, defined as:
  - End-of-TP2 eGFR that is < 90% of the End-of-TP1 eGFR for subjects whose End-of-TP1 eGFR (mean of Week 11 and Week 12 eGFR) is  $\ge 100\%$  of baseline;

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

- o End-of-TP2 eGFR that is < 90% of baseline for subjects whose End-of-TP1 eGFR is  $\ge 90\%$  of baseline and < 100% of baseline.
- Allograft failure (defined by allograft nephrectomy, or institution of permanent dialysis, or return to the transplant waitlist for renal transplant, whichever occurs first)
- Subject death by any cause.

#### All-Cause Allograft Failure

All-cause allograft failure within 48 months after enrollment is defined as 1 of the following, whichever occurs first:

- Allograft failure (defined by allograft nephrectomy, or institution of permanent dialysis, or return to the transplant waitlist for renal transplant, whichever occurs first), OR
- Subject death by any cause.

No subject has reached 48 months after enrollment due to study termination.

#### 8.3 Study Periods Relative to Treatment

#### **8.3.1** Time in Relation to Treatment

Safety data (AEs and concomitant medications) will be assigned to the study time periods defined below (refer to Section 8.1.2 for imputation of incomplete or missing dates).

**Before-therapy** is defined as the date/time prior to the first start of subject's infusion with study treatment.

**On-therapy** is defined as the time from the first start of an infusion of study treatment in Treatment Period 1 up to 30 days after last study drug administration in Treatment Period 2. If a subject had a Retreatment Period, the time still on drug in Retreatment Period (extended to +30 days after last drug in Retreatment Period) will be accounted as On-therapy. In case a subject has more than one Retreatment Periods, the time between Retreatment Periods will be accounted for Follow-up.

**Follow-up** is defined as any time after last study drug administration in Treatment Period 2 plus 30 days. Time of Retreatment Periods are to be excluded from Follow-up, please refer to Ontherapy.

## 8.3.2 Study Time Periods for AEs

AEs occurring On-Therapy or during Follow-up will be handled as treatment-emergent AEs.

Protocol Number: CSL842 3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

## 8.3.3 Study Time Periods for Prior and Concomitant Medications

Prior medications are those ending in the before-therapy period.

Concomitant medications include those that start during the before-therapy period and continue into the on-therapy and Follow-up periods as well as those that start during the on-therapy and Follow-up time periods. Therapies that start during the before-therapy period and have a missing end date will be assumed to continue into the on-therapy period and, therefore, will also be considered concomitant medications.

## 9 Study Population

Only data of subjects who provided informed consent (informed consent date available in the database) will be included in the statistical analysis.

Unless otherwise stated, all tables and listings in this section will be based on the mITT and / or Safety Analysis Set, and all summaries and data listings will use treatment descriptors as specified in Section 7.2.

## 9.1 Disposition of Subjects

The following summaries will be provided by treatment group and for the Screened Analysis Set, as appropriate:

Subject disposition presenting the number and percentages of:

- subjects screened,
- subjects ineligible/failed screening,
- reason for screening failure,
- subjects eligible for Treatment Period 1,
- subjects treated with open-label study medication in Treatment Period 1,
- subjects completed Treatment Period 1,
- subjects discontinued during Treatment Period 1 (before Week 13) and reasons for discontinuation,
- subjects eligible for randomization in Treatment Period 2 (subjects reached week 13 and responded to treatment in Treatment Period 1),
- subjects randomized,
- subjects treated with blinded study medication during Treatment Period 2,
- subjects completed Treatment Period 2,

- subjects discontinued during Treatment Period 2 (before Week 38) and reasons for discontinuation,
- Subjects discontinued from study before week 208,
- subjects available by visit (Treatment Period 1, Treatment Period 2), a subject will be considered to have attended a visit if a visit date is recorded (provided for RiS Analysis Set and RWS Analysis Set).

Number and percentage of subjects in the following analysis sets will be presented:

- Screened Analysis Set,
- Enrolled Analysis Set,
- RiS Analysis Set,
- RWS Analysis Set,
- mITT Analysis Set,
- PK Analysis Set,
- CCI

Number and percentage of subjects in the following categories will be presented:

- Subjects applicable to original protocol,
- Subjects applicable to amendment 1,
- Subjects applicable to amendment 2,
- Subjects applicable to amendment 3.

Reasons for study withdrawal will be presented in the order they are displayed in the eCRF.

A listing will be provided including date of informed consent, date of randomization, date of first treatment (Treatment Period 1, Treatment Period 2, Retreatment Period[s]), study completion, reason if not completed, and assignment to analysis sets.

#### 9.2 Protocol Deviations

The following listings will be provided for the Enrolled Analysis Set:

- All inclusion / exclusion and major protocol deviations.
- All other protocol deviations.

#### 9.3 Demographic and Baseline Characteristics

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

## 9.3.1 Demographics

The following demographic characteristics will be summarized using descriptive statistics or frequency counts, as appropriate:

- Age,
- Age group (< 65 years and  $\ge$ 65 years),
- Sex,
- Ethnicity,
- Race and racial combinations,
- Height,
- Weight,
- BMI,
- Diagnosis of HIV,
- Diagnosis of HBV,
- Diagnosis of HCV.

The weight to be summarized as part of demographics will be the dry weight based on medical history. If the dry weight is missing, the weight at Screening will be used. If the weight at Screening is missing, the Day 1 weight will be used. Demographics will be summarized for the RWS Analysis Set and overall and for RiS Analysis Set.

#### 9.3.2 Baseline Characteristics

The following will be summarized using descriptive statistics or frequency counts, as appropriate:

- Allograft / allograft donor characteristics,
- Diagnosis and disease characteristics.

Baseline characteristics will be summarized for the RWS Analysis Set and overall and for RiS Analysis Set.

 Allograft / allograft donor characteristics: age, sex, ethnicity, race, biological relative, blood group, status at time of donation (alive, dead), deceased donor donation type (donation after brain death, donation after circulatory death), deceased donor criteria (kidney standard criteria donor, kidney expanded criteria donor), Kidney Donor Profile

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

- Index (KDPI score), Human Immunodeficiency Virus (HIV) (yes, no), Hepatitis B Virus (HBV) (yes, no), Hepatitis C Virus (HCV) (yes, no),
- Diagnosis and disease characteristics: time since most recent renal transplant, time since AMR diagnosis, time since most recent rejection episode, severity of current AMR episode, total number of renal transplants, primary reason for kidney transplant (diabetes [type 1 and 2], hypertension, polycystic kidney disease, drug toxicity [non-steroidal anti-inflammatory drugs or others], IgA nephropathy, rapidly progressive neuropathy, membranous glomerulopathy, other nephritides, renal artery stenosis, other infectious diseases [HIV; hepatitis; endotoxin], congenital nephropathy [primary NOS], stone disease, renal cancer, other), delayed graft function (yes, no), dialysis within 14 days after most recent transplant (yes, no), presence of DSA prior to kidney transplant (yes, no), de novo DSA post-transplant (yes, no).

The following listings will be provided for RWS Analysis Set and overall and for RiS Analysis Set:

- Demographic characteristics,
- Allograft / allograft donor characteristics,
- Diagnosis and disease characteristics.

#### 9.4 Prior and Concomitant Medications

Prior and Concomitant medications will be coded using CSL Behring Drug coding dictionary (WHO-DDE Enhanced 2016MAR, B2 Format), summarized, and listed. The summary of prior and concomitant medications will show the number and percentage of subjects taking prior/concomitant medications. Anatomical Therapeutic Chemical (ATC) classification Level 1 (Body System) information will be included in the dataset created but will not appear on the listing or summary. ATC Level 4 and preferred term of prior/concomitant medications will be used for summaries and listings. If the ATC Level 4 coding is not available for a preferred term, the next available lower level ATC code will be used. The summary will be provided by treatment group for RWS Analysis Set and overall for the RiS Analysis Set.

Concomitant medication start and end dates relative to treatment start and end dates are used to select data to include in summaries as follows:

• Summary of Concomitant Medications: This summary will contain medications with start dates relative to treatment assigned to ('BEFORE', 'DURING') and end dates relative to treatment assigned to ('DURING', 'AFTER').

Protocol Number: CSL842 3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

• Summary of Concomitant Medications with On-Therapy Onset: This summary will contain medications with start dates relative to treatment assigned ('DURING') and end dates relative to treatment assigned to ('DURING', 'AFTER').

In the summary of concomitant medications, each subject is counted once within each unique term. For example, if a subject takes Amoxycillin on two separate occasions, the subject is counted only once under the ingredient "Amoxycillin".

Concomitant medications will be summarized separately for medications with onset date within the on-therapy period and for medications with onset date within the before-therapy period.

Note: In order to be considered a concomitant medication, the concomitant medication must have been taken at some point during the on-therapy window.

Concomitant medications will be summarized for the RWS Analysis Set and overall and for RiS Analysis Set.

## 9.5 Medical History

Medical history by body system will be summarized in a frequency table by treatment group for RWS Analysis Set and overall and for RiS Analysis Set.

Medical history will also be presented in a by-subject listing for RiS Analysis Set.

## 10 Efficacy

All efficacy summary will be based on mITT Analysis Set of subjects for Period 2 unless otherwise specified. All efficacy summary will be based on RiS Analysis Set for Period 1 unless otherwise specified.

Subject listings will be provided for the efficacy information based on the mITT Analysis Set.

## 10.1 Analysis of Proportion of Subjects With Loss of Response at the Endof-TP2

The number and proportion of subjects with loss of response at the End-of-TP2 will be presented by treatment group along with the confidence interval for the difference between the two groups.

Subjects will be considered to have lost response if they drop-out or are lost to follow-up before the response status at the End-of-TP2 could be determined.

Components of loss-of-response at the End-of-TP2 will be summarized by treatment groups in terms of the proportion of subjects with:

- End-of-TP2 eGFR (mean of Week 36 and Week 38 eGFR values) that is not stable, defined as:
  - End-of-TP2 eGFR that is < 90% of the End-of-TP1 eGFR for subjects whose End-of-TP1 eGFR is  $\ge 100\%$  of baseline,
  - End-of-TP2 eGFR that is < 90% of baseline for subjects whose End-of-TP1 eGFR is ≥90% of baseline and < 100% of baseline,</li>
- All-cause allograft failure (ie, allograft nephrectomy, or institution of permanent dialysis, or return to the transplant waitlist for renal transplant),
- Death by any cause.

The primary efficacy analysis will be conducted for the mITT Analysis Set.

## 10.1.1 Subgroup Analyses of Proportion of Subjects With Loss of Response at the End-of-TP2

The proportion of subjects with loss of response at the End-of-TP2 will be summarized by the treatment group for the following subgroups based on the following subgroup analyses outlined below will be conducted for the mITT Analysis Set.

The following subgroups, and possibly others to be described in the SAP, will be summarized by treatment group with respect to the proportion of loss-of-response:

- Geographic region: USA, non-USA,
- DSA by randomization strata: sensitized, de novo,
- DSA by classification: HLA class I, HLA class II, both HLA class I and II,
- AMR severity: severe, non-severe (all other severities),
- Type of donor: deceased, living,
- Recipient race: Black, non-Black,
- Recipient sex: Male, Female,
- Recipient age: < 65 years,  $\ge 65$  years.

The difference in the proportion of response along with the 95% confidence interval will be also presented for each subgroup.

Protocol Number: CSL842 3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

## 10.2 Analysis of key Secondary Endpoint Proportion of Subjects With All-Cause Allograft Failure Through the Responder Follow-up Period (ie, Within 48 Months After Enrollment)

No subject will complete the follow-up period of 48 months after enrollment. Therefore, this key secondary analyses cannot be conducted.

## 10.3 Analysis of Time to All-Cause Allograft Failure Through 48 Months After Enrollment

No formal analysis will be conducted for time to all-cause allograft failure since no subject will complete 48 months after enrollment.

A by-listing of all-cause allograft failure information will be provided for the mITT Analysis Set.

## 10.4 Analysis of the Change in eGFR From Baseline to End-of-TP1

This analysis will be based on the RiS Analysis Set.

The eGFRs during Treatment Period 1 (ie with open-label C1-INH) will be summarized by scheduled visit using descriptive statistics for the observed values, and changes from baseline (ie missing data will be not imputed).

## 10.5 Analysis of Responders at the End-of-TP1

This analysis will be based on the RiS Analysis Set.

The proportion of responders at the End-of-TP1 will be presented together with an exact 95% confidence interval. Definition of response at End-of-TP1 is given in Section 8.2.9.

## 10.6 Analysis of the Change in eGFR From End-of-TP1 to the End-of-TP2

No formal analysis for the change in eGFR from End-of-TP1 to the End-of-TP2 will be conducted.

A by-listing for eGFR of all individual values will be provided. for the mITT Analysis Set.

## 10.7 Analysis of the Rate of Change of eGFR in Treatment Period 2

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

No formal analysis of the rate of change of eGFR in Treatment Period 2 will be conducted due to the small number of subjects completing TP2. Mean plot for the change in eGFR from baseline in Treatment Period 2 will be provided for the subjects in the mITT Analysis Set.



#### 10.10 Analysis of C1-INH Functional Activity

PK parameter of  $C_{max}$  and  $AUC_{0-t}$  for C1-INH functional activity will be presented in a bysubject listing for the PK Analysis Set (see Section 12).



## 10.12 Analysis of Plasmapheresis Sessions

The total number plasmapheresis sessions will be derived for each subject and provided in a bylisting for the mITT Analysis Set.



## 10.18 Trough IVIg Concentrations at Designated Time Points

A by-listing of trough IVIg concentrations at will be presented for the RiS Analysis Set at Week 12 and for the mITT Analysis Set at Week 32.

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)



#### 10.20 Treatment Compliance

Percentage compliance will be a function of the amount of IMP taken, ie, the actual cumulative administered volume (mL), and the amount of IMP prescribed, ie, the cumulative planned volume (mL).

Percentage compliance to IMP will be calculated as:

compliance (%) = (cumulative administered volume / cumulative planned volume)\*100.

Percentage compliance will be summarized by frequencies of < 80%, 80% - 120%, > 120%.

Percentage compliance will be summarized for the RiS Analysis Set for Treatment Period 1 and by treatment group for the mITT Analysis Set for Treatment Period 2. Percentage compliance will be also summarized for the entire study for the mITT subjects randomized to C1-INH in period 2. Also, compliance will be summarized based on intravenous delivery and subcutaneous delivery of C1-INH during Treatment Period 1.

Subjects may undergo retreatment during the post-treatment Follow-up Period with the blinded investigational product to which they were randomized in Treatment Period 2.

The following listings will be provided:

- Randomized and actual treatments,
- Drug accountability data (dispensed and returned),
- Overall compliance.

A by-subject listing will be provided including compliance by treatment period, by delivery system (intravenous and subcutaneous), randomized and actual treatments.

Calculation of compliance and extend of exposure (see Section 11.1) will be based on drug accountability data collected by IRT system (or RAVE) as the eCRF does not contain any such related data fields. Drug accountability data will be part of final study data base.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

## 11 Safety Analyses

Open-label safety events and findings will be defined as those with an onset date prior to the randomization date. Double-blind safety events and findings will be defined as those with an onset date on or after the randomization date.

The RiS Analysis Set will be used for analysis of safety for open label TP1. The RWS Analysis Set will be used for analysis of safety during the double-blind period; summaries will be presented by treatment group and total number of subjects in RWS Analysis Set. Also, safety of RWS subjects randomized to C1-INH will be summarized over the study including periods 1 and 2 and follow-up.

## 11.1 Extent of Exposure

The extent of exposure to C1-INH in open-label and in double-blind period and to placebo in double-blind period will be summarized using descriptive statistics. Extent of exposure will be described in terms of the following (including intravenous administration and subcutaneous administrations):

- Cumulative administered volume (mL), calculated as sum of single administered volumes in treatment periods,
- Cumulative planned volume (mL), calculated as sum of single planned volumes in treatment periods (planned administration at days 1, 4, 7, 10, and 13 and twice weekly dosing beginning at the day 14 visit in Treatment Period 1 and twice weekly dosing in Treatment Period 2; dosing scheme must be taken into account for cumulative planned dose depending on subjects time in study; the number of administrations in period of twice weekly dosing will be calculated as: ((date of end of twice weekly dosing date of start of twice weekly dosing +1) / 7) \*2,
- Days on treatment, calculated as days between first and last dose in treatment periods;
- Average daily dose, calculated as cumulative administered dose divided by days on treatment for each treatment period,
- For subjects continuing C1-INH in Treatment Period 2 cumulative administered dose, cumulative planned dose, days on treatment and average daily dose will be summarized for the whole C1-INH treatment period.

Extent of exposure for Retreatment Periods will be summarized separately.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

For summaries of Treatment Period 1 the RiS Analysis Set will be used. Summaries for Treatment Period 2 will be based on the RWS Analysis Set. Also, exposure summary will be presented for the RWS subjects receiving C1-INH during the entire study (Treatment Period 1 and Treatment Period 2 combined).

A by-subject listing will be provided including treatment period (including re-treatment), cumulative administered volume, cumulative planned volume, days on treatment and average daily dose.

#### 11.2 Adverse Events

Adverse events will be coded to the Preferred Term (PT) level using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary), version 23.0 or higher. Treatment-emergent AEs (TEAEs) are defined as AEs reported at or after the start of the first infusion. All AEs regardless of when they were reported will be listed.

Summaries of TEAEs will count the number of subjects, not the number of events, that is, subjects with multiple occurrences of the same TEAE will be counted once.

The number and percentage of subjects with TEAEs will be reported. Also, the number and percentage of subjects with serious TEAEs, TEAEs by severity, and serious TEAEs related to investigational product will be presented. Adverse events will be presented for Treatment Period 1 and RiS Analysis Set. For Treatment Period 2 summaries will be presented for the RWS Analysis Set. In addition, the summaries will be given for C1-INH over the whole study for RWS Analysis Set and a summary across the whole study will be given for the RiS Analysis Set.

A summary of number and percentage of subjects with any TEAE by maximum severity or grade will be produced. TEAEs will be sorted by System Organ Class (SOC) and PT in descending order of incidence overall treatment arms. The summary will report the number of subjects with at least one TEAE, counted for the maximum severity and, for each PT reported, the number of subjects for each, counted for the maximum severity.

In addition, the frequency and percentage of TEAEs will be summarized and displayed in two ways: 1) in descending order of incidence in whole study for RiS Analysis Set by PT only and 2) in descending order of incidence whole study for RiS Analysis Set by SOC and PT. In the SOC row, the number of subjects with multiple events under the same system organ class will be counted once.

A separate summary will be provided for study treatment-related serious TEAEs. Missing relationship to study treatment will be imputed as described in Section 8.1.2; this summary will also include the number and percentage of TEAEs with a missing relationship to aid in interpretation of the results.

By-subject listings will also be provided with detailed information to support the different AE summaries.

## 11.3 Adverse Events of Special Interest (AESI)

Adverse events of special interest of Treatment Period 2 will be presented for the RWS Analysis Set. In addition, adverse events of special interest will be summarized for C1-INH over the whole study for RWS Analysis Set and a summary across the whole study will be given for the RiS Analysis Set.

- Thromboembolic events
  - Systemic thrombotic or thromboembolic events not including catheter or dialysis related clots are of interest. Identification will be based on the Standardized MedDRA Query (SMQ) Embolic and thrombotic events (narrow),
- Anaphylaxis
  - o Anaphylaxis will be identified using the SMQ Anaphylactic reaction (broad).

Treatment-emergent adverse events of special interest will be summarized by SOC and PT.

A separate by-subject listing will be produced for all treatment-emergent adverse events of special interest based on RiS Analysis Set. A listing of terms included in each SMQ can be found in Section 16.1 and 16.2.

#### 11.4 Deaths and Serious Adverse Events

A by-listing will be generated to provide subject-specific details on subjects who died.

The following summaries will be provided for Treatment Period 2 and the RWS Analysis Set. In addition, a summary for C1-INH over the whole study for RWS Analysis Set and a summary across the whole study will be given for the RiS Analysis Set:

• Serious TEAEs,

Serious TEAEs related to Study Treatment.

The following listings will be provided for RiS Analysis Set:

- Serious Non-TEAEs,
- Serious TEAEs,
- TEAEs resulting in death.

## 11.5 Adverse Events Leading to Discontinuation of Study Treatment, Withdrawal from the Study, and Other Significant Adverse Events

The following listings will be provided based on RiS Analysis Set:

- TEAEs Leading to Discontinuation of Study Treatment,
- Non-TEAEs leading to Withdrawal from the Study,
- TEAEs leading to Withdrawal from the Study.

#### 11.6 Pregnancies

While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE or SAE as described in the protocol. If any subject OR any subject or subject's partner becomes pregnant while on the study, the information will be included in the narratives and no separate table or listing will be produced.

#### 11.7 Clinical Laboratory Evaluations

#### 11.7.1 Clinical chemistry

All clinical chemistry parameters for this study will be summarized by scheduled visit using descriptive statistics. All unscheduled visits will be excluded from these by-visit summaries.

Open-label clinical chemistry data for Period 1 and that for the entire study will be summarized for the RiS Analysis Set. Double-blind clinical chemistry data for Period 2 will be summarized for the RWS Analysis Set by treatment.

The estimated and CCI eGFR will be summarized as part of efficacy, and not part of safety.

<u>Clinical Chemistry parameter to be summarized:</u> Albumin, alkaline phosphatase, ALT, AST, total bilirubin, BUN, calcium, carbon dioxide, chloride, creatinine, glucose, potassium, sodium, and protein (total).

## 11.7.2 Hematology

All hematology parameters for this study will be summarized by scheduled visit using descriptive statistics. All unscheduled visits will be excluded from these by-visit summaries.

Open-label hematology data and that for the entire study will be summarized for the RiS Analysis Set.

Double-blind hematology data will be summarized for the RWS Analysis Set by treatment.

Hematology parameter to be summarized: Hemoglobin, hematocrit, red blood cell indices: mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean corpuscular volume, blood cell counts: basophils, eosinophils, erythrocytes, leukocytes, lymphocytes, monocytes, neutrophils, neutrophil band forms, platelets, and reticulocytes.

**DSA:** will be included as efficacy endpoint and will therefore be summarized for efficacy.

## 11.8 Other Safety Measures

## 11.8.1 Vital Signs

Systolic blood pressure, diastolic blood pressure, heart rate, and weight will be summarized for each scheduled visit using descriptive statistics or frequency counts as appropriate.

Vital signs during Treatment Period 1 will be summarized for the RiS Analysis Set. Vital signs for the entire study will be summarized for the RWS Analysis Set by treatment.

#### 12 Pharmacokinetics

All non-compartmental analyses for the derivation of PK parameters will be performed according to CSL SOP PK-GDL-01 and will be performed by CSL Behring Clinical Pharmacology & Pharmacometrics or their designate by using WinNonlin® version 8.1 or later.

All analyses in this section will be based on the PK population, unless otherwise stated.

The merge of PK concentration data and CRF data to generate a dataset with actual blood sampling times, nominal sampling times, actual time relative to dosing, and PK concentrations of

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

C1-INH antigen concentrations and C1-INH functional activity will be performed after data base lock by PPD and is specified in Section 12.5.

#### 12.1 PK Sampling Schedule

Blood samples will be taken for measurement of C1-INH antigen concentrations and C1-INH functional activity at the following time points of Day 10 of Treatment Period 1: pre-dose, 0 minutes (start of C1-INH infusion), 15 minutes, 3, 8, 24, and 72 hours after start of infusion and at Week 11 visit (Treatment Period 1) at time points of: pre-dose, 0 minutes (time of C1-INH injection), 24, 48, and 72 hours after injection. PK samples will be drawn in a subset of subjects. Summary statistics will be provided by nominal (planned) time points.

Concentration data excluded from the derivation of PK parameters will be omitted from summaries and will be flagged with an asterisk in the relevant data listings, with a footnote to indicate that these values have been omitted from subsequent analyses.

### 12.2 Plasma PK Endpoints

The PK parameters based on data collected on Day 10 following IV administration and Week 10 following SC administration will be derived, using Phoenix WinNonlin, Version 8.1 or higher. The PK parameter derivation is based on actual sampling times and includes imputation of the values below the lower limit of quantification (BLQ) and missing data will be conducted in accordance to CSL SOP PK-GDL-01, Guideline on the Conduct of Non-compartmental Pharmacokinetic Analyses, CSL Behring which gives guidance on how to derive PK parameters in the presence of missing data.

Definition of derived PK Parameter:

| Term | Definition |
|---|---|
| AUC <sub>0-t</sub> | Area under the concentration time curve from time point zero to the last quantifiable time point. |
| C <sub>max</sub> | The maximum (peak) observed C1-INH level. |
| $T_{max}$ | The time to reach C <sub>max</sub> . |

Protocol Number: CSL842\_3001

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

| Term | Definition |
|---------------------|------------------------------------------------------|
| C <sub>trough</sub> | Trough C1-INH, collected prior to the next infusion. |

# 12.3 Summary of C1-INH Antigen and Functional Activity Plasma Concentrations

The handling and imputation of BLQ values for PK parameters derivation is described in PK-GDL-01, Guideline on the Conduct of Non-compartmental Pharmacokinetic Analyses, CSL Behring. The imputation rules below will be used for summary statistics of C1-INH antigen and functional activity plasma concentrations. The summaries will be given by sampling time point (planned time points) and treatment group for the PK Analysis Set.

- The sampling time of pre-dose samples relative to dosing will be set to zero.
- Any BLQ in the listing of individual concentrations will be set to missing.
- Set any pre-dose BLQ to zero for summaries.
- Set any BLQ occurring in the profile or at the end of the profile to missing and exclude missing values from the calculation of the means.
- Calculate mean concentrations at any individual time point if at least 50% of the individual values are available (ie are quantifiable and not missing) at this time point otherwise report as "not calculated (NC)".

Summary statistics for concentration-time data will include number of observations, mean, standard deviation, coefficient of variation (CV)%, minimum, median and maximum.

A by-subject listing of C1-INH antigen and functional activity plasma concentration data will support the summaries.

## 12.4 Summary of C1-INH PK Parameters

PK parameters of  $C_{max}$ ,  $AUC_{0-t}$ ,  $C_{trough}$  and for C1-INH antigen and functional activity will be summarized by treatment group for the PK Analysis Set by descriptive statistics with parameter of n, arithmetic mean, SD, CV% (CV% = 100\* standard deviation / mean), minimum, Q25, median, Q75, and maximum.

T<sub>max</sub> will be summarized by descriptive statistics with parameter of n, minimum, Q25, median, Q75, and maximum.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

A by-subject listing of C1-INH PK parameters will be provided.

#### 12.5 Pharmacokinetic Analysis Data Flow

After database lock, PPD will produce the SDTM domains. Domain PC will contain the C1-INH antigen concentrations and C1-INH functional activity concentrations. The PC domain along with domains VS, DM and EX will be provided by PPD . PPD Early Phase Services will derive the PK parameters and produce the PK parameter dataset in Excel format. From this, PPD will produce the SDTM domain PP and eventually the analysis dataset.

Before database lock, PPD will use dummy data for the PK parameters in domain PP to be able to pre-program the planned output.



#### 15 References

Fleiss JL, Levin B, Paik MC. Statistical methods for rates and proportions. 3rd rev. ed. New York: Wiley; 2003.

Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. Erratum in: Ann Intern Med. 2008 Oct 7;149(7):519.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

Loupy A, Haas M, Solez K, Racusen L, Glotz D, Seron D, Nankivell BJ, Colvin RB, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell L, Drachenberg C, Dragun D, de Kort H, Gibson IW, Kraus ES, Lefaucheur C, Legendre C, Liapis H, Muthukumar T, Nickeleit V, Orandi B, Park W, Rabant M, Randhawa P, Reed EF, Roufosse C, Seshan SV, Sis B, Singh HK, Schinstock C, Tambur A, Zeevi A, Mengel M. The Banff 2015 Kidney Meeting Report: Current Challenges in Rejection Classification and Prospects for Adopting Molecular Pathology. Am J Transplant.2017 Jan;17(1):28-41.

Viglietti D, Gosset C, Loupy A, Deville L, Verine J, Zeevi A, Glotz D, Lefaucheur C. C1-inhibitor in Acute Antibody-mediated Rejection Nonresponsive to Conventional Therapy in Kidney Transplant Recipients: A Pilot Study. Am J Transplant. 2016; 16: 1596-1603.

Viglietti D, Loupy A, Duong Van Huyen J, Verine J, Zeevi A, Legendre C, Glotz D, Lefaucheur C. Composite Score to Define the Risk of Allograft Loss After Standard-of-Care Treatement of Antibody-Mediated Rejection in Kidney Transplantation. Am J Transplant. 2016; 16 (Suppl 3).

Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES, Published: November 27, 2017.

PK-GDL-01, Guideline on the Conduct of Non-compartmental Pharmacokinetic Analyses, CSL Behring.

Product Name: C1-esterase Inhibitor, Human (500 IU/mL)

## 16 Appendices

# 16.1 Standardized MedDRA Query for Embolic and Thrombotic Events (Narrow) (SMQ Code: 20000081)

| SMQ Name: Embolic and thrombotic events, arterial (SMQ) | | | | e:20000082 |
|---|---|---|---|---|
| Preferred Term | Code | Level | Scope | Category |
| Acute aortic syndrome | 10074337 | PT | Narrow | A |
| Acute myocardial infarction | 10000891 | PT | Narrow | A |
| Amaurosis | 10001902 | PT | Narrow | A |
| Amaurosis fugax | 10001903 | PT | Narrow | A |
| Angioplasty | 10002475 | PT | Narrow | A |
| Aortic bypass | 10057617 | PT | Narrow | A |
| Aortic embolus | 10002897 | PT | Narrow | A |
| Aortic surgery | 10061651 | PT | Narrow | A |
| Aortic thrombosis | 10002910 | PT | Narrow | A |
| Aortogram abnormal | 10057794 | PT | Narrow | A |
| Arterectomy | 10071026 | PT | Narrow | A |
| Arterectomy with graft replacement | 10003140 | PT | Narrow | A |
| Arterial angioplasty | 10081731 | PT | Narrow | A |
| Arterial bypass occlusion | 10077766 | PT | Narrow | A |
| Arterial bypass operation | 10056418 | PT | Narrow | A |
| Arterial bypass thrombosis | 10077765 | PT | Narrow | A |
| Arterial graft | 10061655 | PT | Narrow | A |
| Arterial occlusive disease | 10062599 | PT | Narrow | A |
| Arterial revascularisation | 10084482 | PT | Narrow | A |
| Arterial stent insertion | 10061657 | PT | Narrow | A |
| Arterial therapeutic procedure | 10052949 | PT | Narrow | A |
| Arterial thrombosis | 10003178 | PT | Narrow | A |
| Arteriogram abnormal | 10061659 | PT | Narrow | A |
| Arteriogram carotid abnormal | 10003195 | PT | Narrow | A |
| Arteriotomy | 10078636 | PT | Narrow | A |
| Atherectomy | 10063025 | PT | Narrow | A |
| Atherosclerotic plaque rupture | 10076604 | PT | Narrow | A |
| Atrial appendage closure | 10079735 | PT | Narrow | A |
| Atrial appendage resection | 10080843 | PT | Narrow | A |
| Basal ganglia infarction | 10069020 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|-----------------------------------|----------|-------|--------|----------|
| Basilar artery occlusion | 10048963 | PT | Narrow | A |
| Basilar artery thrombosis | 10063093 | PT | Narrow | A |
| Blindness transient | 10005184 | PT | Narrow | A |
| Brachiocephalic artery occlusion | 10069694 | PT | Narrow | A |
| Capsular warning syndrome | 10067744 | PT | Narrow | A |
| Carotid angioplasty | 10071260 | PT | Narrow | A |
| Carotid arterial embolus | 10007684 | PT | Narrow | A |
| Carotid artery bypass | 10053003 | PT | Narrow | A |
| Carotid artery occlusion | 10048964 | PT | Narrow | A |
| Carotid artery stent insertion | 10066102 | PT | Narrow | A |
| Carotid artery thrombosis | 10007688 | PT | Narrow | A |
| Carotid endarterectomy | 10007692 | PT | Narrow | A |
| Cerebellar artery occlusion | 10053633 | PT | Narrow | A |
| Cerebellar artery thrombosis | 10008023 | PT | Narrow | A |
| Cerebral artery embolism | 10008088 | PT | Narrow | A |
| Cerebral artery occlusion | 10008089 | PT | Narrow | A |
| Cerebral artery stent insertion | 10081893 | PT | Narrow | A |
| Cerebral artery thrombosis | 10008092 | PT | Narrow | A |
| Cerebral hypoperfusion | 10065384 | PT | Narrow | A |
| Cerebrovascular insufficiency | 10058842 | PT | Narrow | A |
| Cerebrovascular stenosis | 10061751 | PT | Narrow | A |
| Coeliac artery occlusion | 10069696 | PT | Narrow | A |
| Coronary angioplasty | 10050329 | PT | Narrow | A |
| Coronary arterial stent insertion | 10052086 | PT | Narrow | A |
| Coronary artery bypass | 10011077 | PT | Narrow | A |
| Coronary artery embolism | 10011084 | PT | Narrow | A |
| Coronary artery occlusion | 10011086 | PT | Narrow | A |
| Coronary artery reocclusion | 10053261 | PT | Narrow | A |
| Coronary artery surgery | 10011090 | PT | Narrow | A |
| Coronary artery thrombosis | 10011091 | PT | Narrow | A |
| Coronary endarterectomy | 10011101 | PT | Narrow | A |
| Coronary revascularisation | 10049887 | PT | Narrow | A |
| Coronary vascular graft occlusion | 10075162 | PT | Narrow | A |
| Embolia cutis medicamentosa | 10058729 | PT | Narrow | A |
| Embolism arterial | 10014513 | PT | Narrow | A |
| Endarterectomy | 10014648 | PT | Narrow | A |
| Femoral artery embolism | 10068365 | PT | Narrow | A |
| Hepatic artery embolism | 10019635 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|---|---|---|---|---|
| Hepatic artery occlusion | 10051991 | PT | Narrow | A |
| Hepatic artery thrombosis | 10019636 | PT | Narrow | A |
| Hypothenar hammer syndrome | 10063518 | PT | Narrow | A |
| Iliac artery embolism | 10021338 | PT | Narrow | A |
| Iliac artery occlusion | 10064601 | PT | Narrow | A |
| Internal capsule infarction | 10083408 | PT | Narrow | A |
| Intra-aortic balloon placement | 10052989 | PT | Narrow | A |
| Intraoperative cerebral artery occlusion | 10056382 | PT | Narrow | A |
| Ischaemic cerebral infarction | 10060840 | PT | Narrow | A |
| Ischaemic stroke | 10061256 | PT | Narrow | A |
| Lacunar infarction | 10051078 | PT | Narrow | A |
| Leriche syndrome | 10024242 | PT | Narrow | A |
| Mesenteric arterial occlusion | 10027394 | PT | Narrow | A |
| Mesenteric arteriosclerosis | 10065560 | PT | Narrow | A |
| Mesenteric artery embolism | 10027395 | PT | Narrow | A |
| Mesenteric artery stenosis | 10027396 | PT | Narrow | A |
| Mesenteric artery stent insertion | 10071261 | PT | Narrow | A |
| Mesenteric artery thrombosis | 10027397 | PT | Narrow | A |
| Myocardial infarction | 10028596 | PT | Narrow | A |
| Myocardial necrosis | 10028602 | PT | Narrow | A |
| Ophthalmic artery thrombosis | 10081144 | PT | Narrow | A |
| Papillary muscle infarction | 10033697 | PT | Narrow | A |
| Penile artery occlusion | 10068035 | PT | Narrow | A |
| Percutaneous coronary intervention | 10065608 | PT | Narrow | A |
| Peripheral arterial occlusive disease | 10062585 | PT | Narrow | A |
| Peripheral arterial reocclusion | 10069379 | PT | Narrow | A |
| Peripheral artery angioplasty | 10057518 | PT | Narrow | A |
| Peripheral artery bypass | 10072561 | PT | Narrow | A |
| Peripheral artery occlusion | 10057525 | PT | Narrow | A |
| Peripheral artery stent insertion | 10072562 | PT | Narrow | A |
| Peripheral artery surgery | 10082470 | PT | Narrow | A |
| Peripheral artery thrombosis | 10072564 | PT | Narrow | A |
| Peripheral embolism | 10061340 | PT | Narrow | A |
| Peripheral endarterectomy | 10072560 | PT | Narrow | A |
| Popliteal artery entrapment syndrome | 10071642 | PT | Narrow | A |
| Post procedural myocardial infarction | 10066592 | PT | Narrow | A |
| Postinfarction angina | 10058144 | PT | Narrow | A |
| Precerebral artery occlusion | 10036511 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|---|---|---|---|---|
| Precerebral artery thrombosis | 10074717 | PT | Narrow | A |
| Profundaplasty | 10078867 | PT | Narrow | A |
| Pulmonary artery occlusion | 10078201 | PT | Narrow | A |
| Pulmonary artery therapeutic procedure | 10063731 | PT | Narrow | A |
| Pulmonary artery thrombosis | 10037340 | PT | Narrow | A |
| Pulmonary endarterectomy | 10072893 | PT | Narrow | A |
| Pulmonary tumour thrombotic microangiopathy | 10079988 | PT | Narrow | A |
| Renal artery angioplasty | 10057493 | PT | Narrow | A |
| Renal artery occlusion | 10048988 | PT | Narrow | A |
| Renal artery thrombosis | 10038380 | PT | Narrow | A |
| Renal embolism | 10063544 | PT | Narrow | A |
| Retinal artery embolism | 10038826 | PT | Narrow | A |
| Retinal artery occlusion | 10038827 | PT | Narrow | A |
| Retinal artery thrombosis | 10038831 | PT | Narrow | A |
| Silent myocardial infarction | 10049768 | PT | Narrow | A |
| Spinal artery embolism | 10049440 | PT | Narrow | A |
| Spinal artery thrombosis | 10071316 | PT | Narrow | A |
| Splenic artery thrombosis | 10074600 | PT | Narrow | A |
| Splenic embolism | 10068677 | PT | Narrow | A |
| Stress cardiomyopathy | 10066286 | PT | Narrow | A |
| Subclavian artery embolism | 10042332 | PT | Narrow | A |
| Subclavian artery occlusion | 10069695 | PT | Narrow | A |
| Subclavian artery thrombosis | 10042334 | PT | Narrow | A |
| Thromboembolectomy | 10064958 | PT | Narrow | A |
| Thrombotic microangiopathy | 10043645 | PT | Narrow | A |
| Thrombotic thrombocytopenic purpura | 10043648 | PT | Narrow | A |
| Transient ischaemic attack | 10044390 | PT | Narrow | A |
| Truncus coeliacus thrombosis | 10062363 | PT | Narrow | A |
| Vascular pseudoaneurysm thrombosis | 10078269 | PT | Narrow | A |
| Vertebral artery occlusion | 10048965 | PT | Narrow | A |
| Vertebral artery thrombosis | 10057777 | PT | Narrow | A |
| Visual acuity reduced transiently | 10047532 | PT | Narrow | A |

| SMQ Name: Embolic and thrombotic events, venous (SMQ) SMQ Code:2 | | | 20000084 | |
|---|---|---|---|---|
| Preferred Term | Code | Level | Scope | Category |
| Aseptic cavernous sinus thrombosis | 10084527 | PT | Narrow | A |
| Axillary vein thrombosis | 10003880 | PT | Narrow | A |
| Brachiocephalic vein occlusion | 10076837 | PT | Narrow | A |
| Brachiocephalic vein thrombosis | 10063363 | PT | Narrow | A |
| Budd-Chiari syndrome | 10006537 | PT | Narrow | A |
| Catheterisation venous | 10052698 | PT | Narrow | A |
| Cavernous sinus thrombosis | 10007830 | PT | Narrow | A |
| Central venous catheterisation | 10053377 | PT | Narrow | A |
| Cerebral venous sinus thrombosis | 10083037 | PT | Narrow | A |
| Cerebral venous thrombosis | 10008138 | PT | Narrow | A |
| Compression garment application | 10079209 | PT | Narrow | A |
| Deep vein thrombosis | 10051055 | PT | Narrow | A |
| Deep vein thrombosis postoperative | 10066881 | PT | Narrow | A |
| Embolism venous | 10014522 | PT | Narrow | A |
| Hepatic vein embolism | 10078810 | PT | Narrow | A |
| Hepatic vein occlusion | 10058991 | PT | Narrow | A |
| Hepatic vein thrombosis | 10019713 | PT | Narrow | A |
| Homans' sign positive | 10051031 | PT | Narrow | A |
| Iliac vein occlusion | 10058992 | PT | Narrow | A |
| Inferior vena cava syndrome | 10070911 | PT | Narrow | A |
| Inferior vena caval occlusion | 10058987 | PT | Narrow | A |
| Jugular vein embolism | 10081850 | PT | Narrow | A |
| Jugular vein occlusion | 10076835 | PT | Narrow | A |
| Jugular vein thrombosis | 10023237 | PT | Narrow | A |
| Mahler sign | 10075428 | PT | Narrow | A |
| May-Thurner syndrome | 10069727 | PT | Narrow | A |
| Mesenteric vein thrombosis | 10027402 | PT | Narrow | A |
| Mesenteric venous occlusion | 10027403 | PT | Narrow | A |
| Obstetrical pulmonary embolism | 10029925 | PT | Narrow | A |
| Obstructive shock | 10073708 | PT | Narrow | A |
| Ophthalmic vein thrombosis | 10074349 | PT | Narrow | A |
| Ovarian vein thrombosis | 10072059 | PT | Narrow | A |
| Paget-Schroetter syndrome | 10050216 | PT | Narrow | A |
| Pelvic venous thrombosis | 10034272 | PT | Narrow | A |
| Penile vein thrombosis | 10034324 | PT | Narrow | A |
| Peripheral vein occlusion | 10083103 | PT | Narrow | A |
| Peripheral vein thrombus extension | 10082853 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|---|---|---|---|---|
| Phlebectomy | 10048874 | PT | Narrow | A |
| Portal vein cavernous transformation | 10073979 | PT | Narrow | A |
| Portal vein embolism | 10082030 | PT | Narrow | A |
| Portal vein occlusion | 10058989 | PT | Narrow | A |
| Portal vein thrombosis | 10036206 | PT | Narrow | A |
| Portosplenomesenteric venous thrombosis | 10077623 | PT | Narrow | A |
| Post procedural pulmonary embolism | 10063909 | PT | Narrow | A |
| Post thrombotic syndrome | 10048591 | PT | Narrow | A |
| Postoperative thrombosis | 10050902 | PT | Narrow | A |
| Postpartum venous thrombosis | 10036300 | PT | Narrow | A |
| Pulmonary embolism | 10037377 | PT | Narrow | A |
| Pulmonary infarction | 10037410 | PT | Narrow | A |
| Pulmonary microemboli | 10037421 | PT | Narrow | A |
| Pulmonary thrombosis | 10037437 | PT | Narrow | A |
| Pulmonary vein occlusion | 10068690 | PT | Narrow | A |
| Pulmonary veno-occlusive disease | 10037458 | PT | Narrow | A |
| Pulmonary venous thrombosis | 10037459 | PT | Narrow | A |
| Renal vein embolism | 10038547 | PT | Narrow | A |
| Renal vein occlusion | 10056293 | PT | Narrow | A |
| Renal vein thrombosis | 10038548 | PT | Narrow | A |
| Retinal vein occlusion | 10038907 | PT | Narrow | A |
| Retinal vein thrombosis | 10038908 | PT | Narrow | A |
| Septic pulmonary embolism | 10083093 | PT | Narrow | A |
| SI QIII TIII pattern | 10068479 | PT | Narrow | A |
| Splenic vein occlusion | 10068122 | PT | Narrow | A |
| Splenic vein thrombosis | 10041659 | PT | Narrow | A |
| Subclavian vein occlusion | 10079164 | PT | Narrow | A |
| Subclavian vein thrombosis | 10049446 | PT | Narrow | A |
| Superior sagittal sinus thrombosis | 10042567 | PT | Narrow | A |
| Superior vena cava occlusion | 10058988 | PT | Narrow | A |
| Superior vena cava syndrome | 10042569 | PT | Narrow | A |
| Thrombophlebitis | 10043570 | PT | Narrow | A |
| Thrombophlebitis migrans | 10043581 | PT | Narrow | A |
| Thrombophlebitis neonatal | 10043586 | PT | Narrow | A |
| Thrombophlebitis superficial | 10043595 | PT | Narrow | A |
| Thrombosed varicose vein | 10043605 | PT | Narrow | A |
| Thrombosis corpora cavernosa | 10067270 | PT | Narrow | A |
| Transverse sinus thrombosis | 10044457 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|--------------------------------|----------|-------|--------|----------|
| Vena cava embolism | 10047193 | PT | Narrow | A |
| Vena cava filter insertion | 10048932 | PT | Narrow | A |
| Vena cava filter removal | 10074397 | PT | Narrow | A |
| Vena cava thrombosis | 10047195 | PT | Narrow | A |
| Venogram abnormal | 10047209 | PT | Narrow | A |
| Venoocclusive disease | 10062173 | PT | Narrow | A |
| Venoocclusive liver disease | 10047216 | PT | Narrow | A |
| Venous angioplasty | 10077826 | PT | Narrow | A |
| Venous occlusion | 10058990 | PT | Narrow | A |
| Venous operation | 10062175 | PT | Narrow | A |
| Venous recanalisation | 10068605 | PT | Narrow | A |
| Venous repair | 10052964 | PT | Narrow | A |
| Venous stent insertion | 10063389 | PT | Narrow | A |
| Venous thrombosis | 10047249 | PT | Narrow | A |
| Venous thrombosis in pregnancy | 10067030 | PT | Narrow | A |
| Venous thrombosis limb | 10061408 | PT | Narrow | A |
| Venous thrombosis neonatal | 10064602 | PT | Narrow | A |
| Visceral venous thrombosis | 10077829 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|--------------------------------------|----------|-------|--------|----------|
| Administration site thrombosis | 10075968 | PT | Narrow | Α |
| Adrenal thrombosis | 10075178 | PT | Narrow | A |
| Angiogram abnormal | 10060956 | PT | Narrow | A |
| Angiogram cerebral abnormal | 10052906 | PT | Narrow | A |
| Angiogram peripheral abnormal | 10057517 | PT | Narrow | A |
| Antiphospholipid syndrome | 10002817 | PT | Narrow | A |
| Application site thrombosis | 10076026 | PT | Narrow | A |
| Arteriovenous fistula occlusion | 10058562 | PT | Narrow | A |
| Arteriovenous fistula thrombosis | 10003192 | PT | Narrow | A |
| Arteriovenous graft thrombosis | 10053182 | PT | Narrow | A |
| Artificial blood vessel occlusion | 10078895 | PT | Narrow | A |
| Atrial thrombosis | 10048632 | PT | Narrow | A |
| Basal ganglia stroke | 10071043 | PT | Narrow | A |
| Bone infarction | 10049824 | PT | Narrow | A |
| Brain stem embolism | 10074422 | PT | Narrow | A |
| Brain stem infarction | 10006147 | PT | Narrow | A |
| Brain stem stroke | 10068644 | PT | Narrow | A |
| Brain stem thrombosis | 10062573 | PT | Narrow | A |
| Cardiac ventricular thrombosis | 10053994 | PT | Narrow | A |
| Catheter site thrombosis | 10079523 | PT | Narrow | A |
| Cerebellar embolism | 10067167 | PT | Narrow | A |
| Cerebellar infarction | 10008034 | PT | Narrow | A |
| Cerebral congestion | 10076929 | PT | Narrow | A |
| Cerebral infarction | 10008118 | PT | Narrow | A |
| Cerebral infarction foetal | 10008119 | PT | Narrow | A |
| Cerebral ischaemia | 10008120 | PT | Narrow | A |
| Cerebral microembolism | 10078311 | PT | Narrow | A |
| Cerebral microinfarction | 10083668 | PT | Narrow | A |
| Cerebral septic infarct | 10070671 | PT | Narrow | A |
| Cerebral thrombosis | 10008132 | PT | Narrow | A |
| Cerebral vascular occlusion | 10076895 | PT | Narrow | A |
| Cerebrospinal thrombotic tamponade | 10052173 | PT | Narrow | A |
| Cerebrovascular accident | 10008190 | PT | Narrow | A |
| Cerebrovascular accident prophylaxis | 10049165 | PT | Narrow | A |
| Cerebrovascular disorder | 10008196 | PT | Narrow | A |
| Cerebrovascular operation | 10051902 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|---|---|---|---|---|
| Choroidal infarction | 10057403 | PT | Narrow | A |
| Collateral circulation | 10069729 | PT | Narrow | A |
| Coronary bypass thrombosis | 10059025 | PT | Narrow | A |
| Device embolisation | 10074896 | PT | Narrow | A |
| Device occlusion | 10064685 | PT | Narrow | A |
| Device related thrombosis | 10077455 | PT | Narrow | A |
| Diplegia | 10013033 | PT | Narrow | A |
| Directional Doppler flow tests abnormal | 10013048 | PT | Narrow | A |
| Disseminated intravascular coagulation | 10013442 | PT | Narrow | A |
| Disseminated intravascular coagulation in newborn | 10013443 | PT | Narrow | A |
| Embolic cerebellar infarction | 10084072 | PT | Narrow | A |
| Embolic cerebral infarction | 10060839 | PT | Narrow | A |
| Embolic pneumonia | 10065680 | PT | Narrow | A |
| Embolic stroke | 10014498 | PT | Narrow | A |
| Embolism | 10061169 | PT | Narrow | A |
| Eye infarction | 10083006 | PT | Narrow | A |
| Fluorescence angiogram abnormal | 10083087 | PT | Narrow | A |
| Foetal cerebrovascular disorder | 10053601 | PT | Narrow | A |
| Gastric infarction | 10084858 | PT | Narrow | A |
| Graft thrombosis | 10051269 | PT | Narrow | A |
| Haemorrhagic adrenal infarction | 10079902 | PT | Narrow | A |
| Haemorrhagic cerebral infarction | 10019005 | PT | Narrow | A |
| Haemorrhagic infarction | 10019013 | PT | Narrow | A |
| Haemorrhagic stroke | 10019016 | PT | Narrow | A |
| Haemorrhagic transformation stroke | 10055677 | PT | Narrow | A |
| Haemorrhoids thrombosed | 10019023 | PT | Narrow | A |
| Hemiparesis | 10019465 | PT | Narrow | A |
| Hemiplegia | 10019468 | PT | Narrow | A |
| Heparin-induced thrombocytopenia | 10062506 | PT | Narrow | A |
| Hepatic infarction | 10019680 | PT | Narrow | A |
| Hepatic vascular thrombosis | 10074494 | PT | Narrow | A |
| Implant site thrombosis | 10063868 | PT | Narrow | A |
| Incision site vessel occlusion | 10076839 | PT | Narrow | A |
| Infarction | 10061216 | PT | Narrow | A |
| Infusion site thrombosis | 10065489 | PT | Narrow | A |
| Injection site thrombosis | 10022104 | PT | Narrow | A |
| Inner ear infarction | 10070754 | PT | Narrow | A |
| Instillation site thrombosis | 10073625 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|-------------------------------------|----------|-------|--------|----------|
| Intestinal infarction | 10022657 | PT | Narrow | A |
| Intracardiac mass | 10066087 | PT | Narrow | A |
| Intracardiac thrombus | 10048620 | PT | Narrow | A |
| Lambl's excrescences | 10083691 | PT | Narrow | A |
| Medical device site thrombosis | 10076145 | PT | Narrow | A |
| Mesenteric vascular insufficiency | 10027401 | PT | Narrow | A |
| Mesenteric vascular occlusion | 10074583 | PT | Narrow | A |
| Microembolism | 10073734 | PT | Narrow | A |
| Monoparesis | 10027925 | PT | Narrow | A |
| Monoplegia | 10027926 | PT | Narrow | A |
| Optic nerve infarction | 10030936 | PT | Narrow | A |
| Pancreatic infarction | 10068239 | PT | Narrow | A |
| Paradoxical embolism | 10066059 | PT | Narrow | A |
| Paraneoplastic thrombosis | 10079251 | PT | Narrow | A |
| Paraparesis | 10033885 | PT | Narrow | A |
| Paraplegia | 10033892 | PT | Narrow | A |
| Paresis | 10033985 | PT | Narrow | A |
| Peripheral revascularisation | 10053351 | PT | Narrow | A |
| Pituitary infarction | 10035092 | PT | Narrow | A |
| Placental infarction | 10064620 | PT | Narrow | A |
| Pneumatic compression therapy | 10059829 | PT | Narrow | A |
| Portal shunt procedure | 10077479 | PT | Narrow | A |
| Post procedural stroke | 10066591 | PT | Narrow | A |
| Postpartum thrombosis | 10077022 | PT | Narrow | A |
| Prosthetic cardiac valve thrombosis | 10063176 | PT | Narrow | A |
| Prosthetic vessel implantation | 10068628 | PT | Narrow | A |
| Quadriparesis | 10049680 | PT | Narrow | A |
| Quadriplegia | 10037714 | PT | Narrow | A |
| Renal infarct | 10038470 | PT | Narrow | A |
| Renal vascular thrombosis | 10072226 | PT | Narrow | A |
| Retinal infarction | 10051742 | PT | Narrow | A |
| Retinal vascular thrombosis | 10062108 | PT | Narrow | A |
| Revascularisation procedure | 10084091 | PT | Narrow | A |
| Shunt occlusion | 10040621 | PT | Narrow | A |
| Shunt thrombosis | 10059054 | PT | Narrow | A |
| Spinal cord infarction | 10058571 | PT | Narrow | A |
| Spinal stroke | 10082031 | PT | Narrow | A |
| Splenic infarction | 10041648 | PT | Narrow | A |

| Preferred Term | Code | Level | Scope | Category |
|---------------------------------|----------|-------|--------|----------|
| Splenic thrombosis | 10074601 | PT | Narrow | A |
| Stoma site thrombosis | 10074515 | PT | Narrow | A |
| Stroke in evolution | 10059613 | PT | Narrow | A |
| Strokectomy | 10084735 | PT | Narrow | A |
| Surgical vascular shunt | 10058408 | PT | Narrow | A |
| Testicular infarction | 10043337 | PT | Narrow | A |
| Thalamic infarction | 10064961 | PT | Narrow | A |
| Thrombectomy | 10043530 | PT | Narrow | A |
| Thromboangiitis obliterans | 10043540 | PT | Narrow | A |
| Thrombolysis | 10043568 | PT | Narrow | A |
| Thrombosis | 10043607 | PT | Narrow | A |
| Thrombosis in device | 10062546 | PT | Narrow | A |
| Thrombosis mesenteric vessel | 10043626 | PT | Narrow | A |
| Thrombosis prophylaxis | 10043634 | PT | Narrow | A |
| Thrombotic cerebral infarction | 10067347 | PT | Narrow | A |
| Thrombotic stroke | 10043647 | PT | Narrow | A |
| Thyroid infarction | 10043742 | PT | Narrow | A |
| Tumour embolism | 10045168 | PT | Narrow | A |
| Tumour thrombectomy | 10081994 | PT | Narrow | A |
| Tumour thrombosis | 10068067 | PT | Narrow | A |
| Ultrasonic angiogram abnormal | 10061604 | PT | Narrow | A |
| Ultrasound Doppler abnormal | 10045413 | PT | Narrow | A |
| Umbilical cord occlusion | 10076714 | PT | Narrow | A |
| Umbilical cord thrombosis | 10071652 | PT | Narrow | A |
| Vaccination site thrombosis | 10076190 | PT | Narrow | A |
| Vascular access site thrombosis | 10078675 | PT | Narrow | A |
| Vascular device occlusion | 10080803 | PT | Narrow | A |
| Vascular graft | 10067740 | PT | Narrow | A |
| Vascular graft occlusion | 10049060 | PT | Narrow | A |
| Vascular graft thrombosis | 10069922 | PT | Narrow | A |
| Vascular operation | 10049071 | PT | Narrow | A |
| Vascular stent insertion | 10063382 | PT | Narrow | A |
| Vascular stent occlusion | 10077143 | PT | Narrow | A |
| Vascular stent thrombosis | 10063934 | PT | Narrow | A |

| Product Name: C1-esterase |
|------------------------------|
| Inhibitor, Human (500 IU/mL) |

| Preferred Term | Code | Level | Scope | Category |
|---|---|---|---|---|
| Vasodilation procedure | 10058794 | PT | Narrow | A |
| Vessel puncture site occlusion | 10076838 | PT | Narrow | A |
| Vessel puncture site thrombosis | 10070649 | PT | Narrow | A |
| Visual midline shift syndrome | 10066856 | PT | Narrow | A |
| SMQ Export: 23.1 - English 2/12/2020 8:42:53 | | | | |
| PM | | | | |

### Standardized MedDRA Query - Anaphylactic Reaction (Broad) (SMQ 16.2 Code: 20000021)

| SMQ Name: Anaphylactic reaction (SMQ) | | | SMQ Cod | SMQ Code: 20000021 |
|---|---|---|---|---|
| Preferred term | Code | Level | Scope | Category |
| Anaphylactic reaction | 10002198 | PT | Narrow | A |
| Anaphylactic shock | 10002199 | PT | Narrow | A |
| Anaphylactic transfusion reaction | 10067113 | PT | Narrow | A |
| Anaphylactoid reaction | 10002216 | PT | Narrow | A |
| Anaphylactoid shock | 10063119 | PT | Narrow | A |
| Circulatory collapse | 10009192 | PT | Narrow | A |
| Dialysis membrane reaction | 10076665 | PT | Narrow | A |
| Kounis syndrome | 10069167 | PT | Narrow | A |
| Procedural shock | 10080894 | PT | Narrow | A |
| Shock | 10040560 | PT | Narrow | A |
| Shock symptom | 10040581 | PT | Narrow | A |
| Type I hypersensitivity | 10045240 | PT | Narrow | A |
| Acute respiratory failure | 10001053 | PT | Broad | В |
| Asthma | 10003553 | PT | Broad | В |
| Bronchial oedema | 10056695 | PT | Broad | В |
| Bronchospasm | 10006482 | PT | Broad | В |
| Cardio-respiratory distress | 10049874 | PT | Broad | В |
| Chest discomfort | 10008469 | PT | Broad | В |
| Choking | 10008589 | PT | Broad | В |
| Choking sensation | 10008590 | PT | Broad | В |
| Circumoral oedema | 10052250 | PT | Broad | В |
| Cough | 10011224 | PT | Broad | В |
| Cough variant asthma | 10063076 | PT | Broad | В |

| Preferred term | Code | Level | Scope | Category |
|----------------------------------|----------|-------|-------|----------|
| Cyanosis | 10011703 | PT | Broad | В |
| Dyspnoea | 10013968 | PT | Broad | В |
| Hyperventilation | 10020910 | PT | Broad | В |
| Irregular breathing | 10076213 | PT | Broad | В |
| Laryngeal dyspnoea | 10052390 | PT | Broad | В |
| Laryngeal oedema | 10023845 | PT | Broad | В |
| Laryngospasm | 10023891 | PT | Broad | В |
| Laryngotracheal oedema | 10023893 | PT | Broad | В |
| Mouth swelling | 10075203 | PT | Broad | В |
| Nasal obstruction | 10028748 | PT | Broad | В |
| Oedema mouth | 10030110 | PT | Broad | В |
| Oropharyngeal oedema | 10078783 | PT | Broad | В |
| Oropharyngeal spasm | 10031111 | PT | Broad | В |
| Oropharyngeal swelling | 10031118 | PT | Broad | В |
| Pharyngeal oedema | 10034829 | PT | Broad | В |
| Pharyngeal swelling | 10082270 | PT | Broad | В |
| Respiratory arrest | 10038669 | PT | Broad | В |
| Respiratory distress | 10038687 | PT | Broad | В |
| Respiratory failure | 10038695 | PT | Broad | В |
| Reversible airways obstruction | 10062109 | PT | Broad | В |
| Sensation of foreign body | 10061549 | PT | Broad | В |
| Sneezing | 10041232 | PT | Broad | В |
| Stridor | 10042241 | PT | Broad | В |
| Swollen tongue | 10042727 | PT | Broad | В |
| Tachypnoea | 10043089 | PT | Broad | В |
| Throat tightness | 10043528 | PT | Broad | В |
| Tongue oedema | 10043967 | PT | Broad | В |
| Tracheal obstruction | 10044291 | PT | Broad | В |
| Tracheal oedema | 10044296 | PT | Broad | В |
| Upper airway obstruction | 10067775 | PT | Broad | В |
| Wheezing | 10047924 | PT | Broad | В |
| Acquired C1 inhibitor deficiency | 10081035 | PT | Broad | С |
| Allergic oedema | 10060934 | PT | Broad | C |
| Angioedema | 10002424 | PT | Broad | С |
| Circumoral swelling | 10081703 | PT | Broad | С |
| Erythema | 10015150 | PT | Broad | С |
| Eye oedema | 10052139 | PT | Broad | С |

| Preferred term | Code | Level | Scope | Category |
|---|---|---|---|---|
| Eye pruritus | 10052140 | PT | Broad | С |
| Eye swelling | 10015967 | PT | Broad | С |
| Eyelid oedema | 10015993 | PT | Broad | С |
| Face oedema | 10016029 | PT | Broad | С |
| Flushing | 10016825 | PT | Broad | С |
| Hereditary angioedema with C1 esterase inhibitor deficiency | 10080955 | PT | Broad | С |
| Injection site urticaria | 10022107 | PT | Broad | C |
| Lip oedema | 10024558 | PT | Broad | C |
| Lip swelling | 10024570 | PT | Broad | C |
| Nodular rash | 10075807 | PT | Broad | С |
| Ocular hyperaemia | 10030041 | PT | Broad | С |
| Oedema | 10030095 | PT | Broad | С |
| Oedema blister | 10080039 | PT | Broad | С |
| Periorbital oedema | 10034545 | PT | Broad | С |
| Periorbital swelling | 10056647 | PT | Broad | С |
| Pruritus | 10037087 | PT | Broad | С |
| Pruritus allergic | 10063438 | PT | Broad | С |
| Rash | 10037844 | PT | Broad | С |
| Rash erythematous | 10037855 | PT | Broad | С |
| Rash pruritic | 10037884 | PT | Broad | С |
| Skin swelling | 10053262 | PT | Broad | C |
| Swelling | 10042674 | PT | Broad | С |
| Swelling face | 10042682 | PT | Broad | C |
| Swelling of eyelid | 10042690 | PT | Broad | С |
| Urticaria | 10046735 | PT | Broad | C |
| Urticaria papular | 10046750 | PT | Broad | С |
| Blood pressure decreased | 10005734 | PT | Broad | D |
| Blood pressure diastolic decreased | 10005737 | PT | Broad | D |
| Blood pressure systolic decreased | 10005758 | PT | Broad | D |
| Cardiac arrest | 10007515 | PT | Broad | D |
| Cardio-respiratory arrest | 10007617 | PT | Broad | D |
| Cardiovascular insufficiency | 10065929 | PT | Broad | D |
| Diastolic hypotension | 10066077 | PT | Broad | D |

| Preferred term | Code | Level | Scope | Category |
|---------------------------------------|----------|-------|-------|----------|
| Hypotension | 10021097 | PT | Broad | D |
| Hypotensive crisis | 10083659 | PT | Broad | D |
| Post procedural hypotension | 10084013 | PT | Broad | D |
| SMQ Export: 23.1 - English (2/12/2020 | | | | |
| 8:39:05 PM) | | | | |

## Signature Page

## CSL842\_3001 - Statistical Analysis Plan - v1 - 10Dec2020

| Signed By | | Date (GMT) |
|--------------|----------|----------------------|
| PPD | | 11-Dec-2020 21:07:52 |
| Approved-PPD | Approval | |
| PPD | | 12-Dec-2020 14:30:23 |
| Approved-PPD | Approval | |
| PPD | | 14-Dec-2020 16:07:05 |
| Approved-PPD | Approval | |

Signature Page 1 of 1

--- Do Not Detach This Signature Page ---

glbdctmp Print Date: 18-Aug-2021 09:52:50 GMT-04:00